CLINICAL TRIAL: NCT00262600
Title: Randomized Evaluation of Long Term Anticoagulant Therapy (RE-LY) Comparing the Efficacy and Safety of Two Blinded Doses of Dabigatran Etexilate With Open Label Warfarin for the Prevention of Stroke and Systemic Embolism in Patients With Non-valvular Atrial Fibrillation: Prospective, Multi-centre, Parallel-group, Non-inferiority Trial (RE-LY Study)
Brief Title: Randomized Evaluation of Long Term Anticoagulant Therapy (RE-LY) With Dabigatran Etexilate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Population Health Research Institute (Other); Uppsala University (Other)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 1160.26; 2005-003894-26 (EudraCT Number: EudraCT)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2011-02-10 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2014-04

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Warfarin

ARMS (3):
- Dabigatran dose 2 (Active Comparator): twice a day
  Interventions: Drug: Dabigatran dose 2
- Warfarin (Active Comparator): once a day
  Interventions: Drug: warfarin
- Dabigatran dose 1 (Active Comparator): twice a day
  Interventions: Drug: Dabigatran dose 1

INTERVENTIONS:
Drug: warfarin — once a day
  Arms: Warfarin
Drug: Dabigatran dose 1 — twice daily
  Arms: Dabigatran dose 1
Drug: Dabigatran dose 2 — twice a day
  Arms: Dabigatran dose 2

SUMMARY:
The primary objective of this trial is to demonstrate the efficacy and safety of dabigatran etexilate in patients with non-valvular atrial fibrillation for the prevention of stroke and systemic embolism.

ELIGIBILITY:
Inclusion criteria Patients with non-valvular atrial fibrillation (AF), at moderate to high risk of stroke, or systemic embolism with at least one additional risk factor (i.e. previous ischemic stroke, TIA, or systemic embolism, left ventricular dysfunction, age >=75 years, age >=65 with either diabetes mellitus, history of coronary artery disease or hypertension)

Exclusion criteria

1. Prosthetic heart valves requiring anticoagulation per se, or hemodynamically relevant valve disease that is expected to require surgical intervention during the course of the study
2. Severe, disabling stroke within the previous 6 months, or any stroke within the previous 14 days
3. Conditions associated with an increased risk of bleeding
4. Contraindication to warfarin treatment
5. Reversible causes of atrial fibrillation (e.g., cardiac surgery, pulmonary embolism, untreated hyperthyroidism).
6. Plan to perform a pulmonary vein ablation or surgery for cure of the AF
7. Severe renal impairment (estimated creatinine clearance <=30 mL/min)
8. Active infective endocarditis
9. Active liver disease
10. Women who are pregnant, lactating, or of childbearing potential who refuse to use a medically acceptable form of contraception throughout the study
11. Anaemia (haemoglobin <100g/L) or thrombocytopenia (platelet count <100 x 109/L)
12. Patients who have developed transaminase elevations upon exposure to ximelagatran
13. Patients who have received an investigational drug in the past 30 days or are participating in another drug study
14. Patients considered unreliable by the investigator concerning the requirements for follow-up during the study and/or compliance with study drug administration, has a life expectancy less than the expected duration of the trial due to concomitant disease, or has any condition which in the opinion of the investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse)
15. Any known hypersensitivity to galactose if the warfarin used contains galactose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18113 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (984):
- United States (374):
  - 1160.26.0009 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.26.0046 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.26.0057 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.26.0211 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.26.0206 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1160.26.0115 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1160.26.0104 Boehringer Ingelheim Investigational Site, Lake Havasu City, Arizona
  - 1160.26.0304 Boehringer Ingelheim Investigational Site, Peoria, Arizona
  - 1160.26.0185 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1160.26.0305 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1160.26.0038 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 1160.26.0302 Boehringer Ingelheim Investigational Site, Jonesboro, Arkansas
  - 1160.26.0121 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.26.0191 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.26.0204 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.26.0213 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.26.0455 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.26.0388 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1160.26.0441 Boehringer Ingelheim Investigational Site, Carmichael, California
  - 1160.26.0145 Boehringer Ingelheim Investigational Site, French Camp, California
  - 1160.26.0333 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 1160.26.0384 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1160.26.0091 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1160.26.0246 Boehringer Ingelheim Investigational Site, Lancaster, California
  - 1160.26.0345 Boehringer Ingelheim Investigational Site, Larkspur, California
  - 1160.26.0217 Boehringer Ingelheim Investigational Site, Loma Linda, California
  - 1160.26.0059 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1160.26.0088 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1160.26.0337 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1160.26.0326 Boehringer Ingelheim Investigational Site, Mather, California
  - 1160.26.0070 Boehringer Ingelheim Investigational Site, Merced, California
  - 1160.26.0349 Boehringer Ingelheim Investigational Site, Oakland, California
  - 1160.26.0016 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1160.26.0087 Boehringer Ingelheim Investigational Site, Palm Springs, California
  - 1160.26.0459 Boehringer Ingelheim Investigational Site, Pasadena, California
  - 1160.26.0216 Boehringer Ingelheim Investigational Site, Redondo Beach, California
  - 1160.26.0135 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1160.26.0162 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1160.26.0300 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1160.26.0371 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1160.26.0116 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1160.26.0148 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1160.26.0270 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1160.26.0284 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1160.26.0351 Boehringer Ingelheim Investigational Site, Santa Ana, California
  - 1160.26.0043 Boehringer Ingelheim Investigational Site, Santa Rosa, California
  - 1160.26.0462 Boehringer Ingelheim Investigational Site, Sylmar, California
  - 1160.26.0276 Boehringer Ingelheim Investigational Site, Torrance, California
  - 1160.26.0379 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1160.26.0419 Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - 1160.26.0321 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1160.26.0449 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1160.26.0360 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1160.26.0413 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1160.26.0362 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1160.26.0399 Boehringer Ingelheim Investigational Site, Greeley, Colorado
  - 1160.26.0058 Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - 1160.26.0241 Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - 1160.26.0278 Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - 1160.26.0085 Boehringer Ingelheim Investigational Site, Fairfield, Connecticut
  - 1160.26.0482 Boehringer Ingelheim Investigational Site, Guilford, Connecticut
  - 1160.26.0366 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 1160.26.0343 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1160.26.0022 Boehringer Ingelheim Investigational Site, Atlantis, Florida
  - 1160.26.0382 Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - 1160.26.0056 Boehringer Ingelheim Investigational Site, Brandon, Florida
  - 1160.26.0105 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.26.0296 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.26.0429 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.26.0376 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 1160.26.0411 Boehringer Ingelheim Investigational Site, Deerfield Beach, Florida
  - 1160.26.0074 Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - 1160.26.0239 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 1160.26.0260 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1160.26.0265 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1160.26.0100 Boehringer Ingelheim Investigational Site, Inverness, Florida
  - 1160.26.0033 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.26.0089 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.26.0232 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.26.0240 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.26.0427 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.26.0464 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.26.0209 Boehringer Ingelheim Investigational Site, Jacksonville Beach, Florida
  - 1160.26.0012 Boehringer Ingelheim Investigational Site, Lakeland, Florida
  - 1160.26.0259 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 1160.26.0358 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 1160.26.0034 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1160.26.0199 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1160.26.0227 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1160.26.0095 Boehringer Ingelheim Investigational Site, Ormond Beach, Florida
  - 1160.26.0037 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1160.26.0076 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1160.26.0081 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1160.26.0111 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1160.26.0137 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1160.26.0389 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1160.26.0417 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1160.26.0332 Boehringer Ingelheim Investigational Site, Rockledge, Florida
  - 1160.26.0226 Boehringer Ingelheim Investigational Site, Safety Harbor, Florida
  - 1160.26.0031 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1160.26.0385 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1160.26.0015 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1160.26.0339 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1160.26.0010 Boehringer Ingelheim Investigational Site, Stuart, Florida
  - 1160.26.0327 Boehringer Ingelheim Investigational Site, Tamarac, Florida
  - 1160.26.0271 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1160.26.0328 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1160.26.0381 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1160.26.0019 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 1160.26.0159 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1160.26.0283 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1160.26.0338 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1160.26.0021 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 1160.26.0319 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 1160.26.0092 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1160.26.0161 Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - 1160.26.0026 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1160.26.0218 Boehringer Ingelheim Investigational Site, Berwyn, Illinois
  - 1160.26.0184 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1160.26.0233 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1160.26.0324 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1160.26.0457 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1160.26.0237 Boehringer Ingelheim Investigational Site, Evanston, Illinois
  - 1160.26.0236 Boehringer Ingelheim Investigational Site, Glenview, Illinois
  - 1160.26.0396 Boehringer Ingelheim Investigational Site, Hines, Illinois
  - 1160.26.0438 Boehringer Ingelheim Investigational Site, Maywood, Illinois
  - 1160.26.0331 Boehringer Ingelheim Investigational Site, Melrose Park, Illinois
  - 1160.26.0364 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 1160.26.0109 Boehringer Ingelheim Investigational Site, North Chicago, Illinois
  - 1160.26.0152 Boehringer Ingelheim Investigational Site, Oak Lawn, Illinois
  - 1160.26.0198 Boehringer Ingelheim Investigational Site, Rockford, Illinois
  - 1160.26.0433 Boehringer Ingelheim Investigational Site, Winfield, Illinois
  - 1160.26.0041 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1160.26.0377 Boehringer Ingelheim Investigational Site, Fort Wayne, Indiana
  - 1160.26.0288 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1160.26.0352 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1160.26.0436 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1160.26.0028 Boehringer Ingelheim Investigational Site, Jeffersonville, Indiana
  - 1160.26.0235 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 1160.26.0268 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 1160.26.0001 Boehringer Ingelheim Investigational Site, West Des Moines, Iowa
  - 1160.26.0189 Boehringer Ingelheim Investigational Site, West Des Moines, Iowa
  - 1160.26.0357 Boehringer Ingelheim Investigational Site, West Des Moines, Iowa
  - 1160.26.0354 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1160.26.0077 Boehringer Ingelheim Investigational Site, Bowling Green, Kentucky
  - 1160.26.0138 Boehringer Ingelheim Investigational Site, Crestview Hills, Kentucky
  - 1160.26.0422 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1160.26.0178 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1160.26.0397 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1160.26.0310 Boehringer Ingelheim Investigational Site, Owensboro, Kentucky
  - 1160.26.0011 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1160.26.0144 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1160.26.0404 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1160.26.0093 Boehringer Ingelheim Investigational Site, Covington, Louisiana
  - 1160.26.0340 Boehringer Ingelheim Investigational Site, Lacombe, Louisiana
  - 1160.26.0018 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1160.26.0391 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1160.26.0252 Boehringer Ingelheim Investigational Site, Morgan City, Louisiana
  - 1160.26.0132 Boehringer Ingelheim Investigational Site, New Iberia, Louisiana
  - 1160.26.0299 Tulane University School Of Medicine, New Orleans, Louisiana
  - 1160.26.0048 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1160.26.0096 Boehringer Ingelheim Investigational Site, Auburn, Maine
  - 1160.26.0068 Boehringer Ingelheim Investigational Site, Scarborough, Maine
  - 1160.26.0114 Boehringer Ingelheim Investigational Site, Annapolis, Maryland
  - 1160.26.0164 Boehringer Ingelheim Investigational Site, Annapolis, Maryland
  - 1160.26.0023 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.26.0047 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.26.0079 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.26.0186 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.26.0194 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.26.0255 Boehringer Ingelheim Investigational Site, Bel Air, Maryland
  - 1160.26.0398 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1160.26.0177 Boehringer Ingelheim Investigational Site, Rockville, Maryland
  - 1160.26.0073 Boehringer Ingelheim Investigational Site, Salisbury, Maryland
  - 1160.26.0207 Boehringer Ingelheim Investigational Site, Salisbury, Maryland
  - 1160.26.0196 Boehringer Ingelheim Investigational Site, Takoma Park, Maryland
  - 1160.26.0187 Boehringer Ingelheim Investigational Site, Towson, Maryland
  - 1160.26.0052 Boehringer Ingelheim Investigational Site, Westminster, Maryland
  - 1160.26.0042 Boehringer Ingelheim Investigational Site, Ayer, Massachusetts
  - 1160.26.0401 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1160.26.0160 Boehringer Ingelheim Investigational Site, East Bridgewater, Massachusetts
  - 1160.26.0443 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 1160.26.0452 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 1160.26.0029 Boehringer Ingelheim Investigational Site, Natick, Massachusetts
  - 1160.26.0446 Boehringer Ingelheim Investigational Site, Newtown, Massachusetts
  - 1160.26.0003 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1160.26.0470 Boehringer Ingelheim Investigational Site, Northborough, Massachusetts
  - 1160.26.0308 Boehringer Ingelheim Investigational Site, Worcester, Massachusetts
  - 1160.26.0141 Boehringer Ingelheim Investigational Site, Bloomfield Hills, Michigan
  - 1160.26.0225 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1160.26.0154 Boehringer Ingelheim Investigational Site, Grand Blanc, Michigan
  - 1160.26.0030 Boehringer Ingelheim Investigational Site, Grand Rapids, Michigan
  - 1160.26.0171 Boehringer Ingelheim Investigational Site, Kalamazoo, Michigan
  - 1160.26.0205 Boehringer Ingelheim Investigational Site, Lapeer, Michigan
  - 1160.26.0279 Boehringer Ingelheim Investigational Site, Muskegon, Michigan
  - 1160.26.0445 Boehringer Ingelheim Investigational Site, Petoskey, Michigan
  - 1160.26.0274 Boehringer Ingelheim Investigational Site, Rochester Hills, Michigan
  - 1160.26.0165 Boehringer Ingelheim Investigational Site, Saginaw, Michigan
  - 1160.26.0020 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 1160.26.0188 Boehringer Ingelheim Investigational Site, Ypsilanti, Michigan
  - 1160.26.0131 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1160.26.0421 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1160.26.0202 Boehringer Ingelheim Investigational Site, Robbinsdale, Minnesota
  - 1160.26.0101 Boehringer Ingelheim Investigational Site, Saint Paul, Minnesota
  - 1160.26.0086 Boehringer Ingelheim Investigational Site, Gulfport, Mississippi
  - 1160.26.0119 Boehringer Ingelheim Investigational Site, Tupelo, Mississippi
  - 1160.26.0055 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 1160.26.0172 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 1160.26.0257 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1160.26.0266 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1160.26.0336 Boehringer Ingelheim Investigational Site, Saint Charles, Missouri
  - 1160.26.0249 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1160.26.0027 Boehringer Ingelheim Investigational Site, Kalispell, Montana
  - 1160.26.0128 Boehringer Ingelheim Investigational Site, Alliance, Nebraska
  - 1160.26.0110 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1160.26.0355 Boehringer Ingelheim Investigational Site, Papillion, Nebraska
  - 1160.26.0346 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1160.26.0066 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1160.26.0174 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1160.26.0430 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1160.26.0190 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 1160.26.0142 Boehringer Ingelheim Investigational Site, Browns Mills, New Jersey
  - 1160.26.0125 Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - 1160.26.0432 Boehringer Ingelheim Investigational Site, Elmer, New Jersey
  - 1160.26.0448 Boehringer Ingelheim Investigational Site, Englewood, New Jersey
  - 1160.26.0248 Boehringer Ingelheim Investigational Site, Flemington, New Jersey
  - 1160.26.0244 Boehringer Ingelheim Investigational Site, Haddon Heights, New Jersey
  - 1160.26.0243 Boehringer Ingelheim Investigational Site, New Brunswick, New Jersey
  - 1160.26.0478 Boehringer Ingelheim Investigational Site, Oakland, New Jersey
  - 1160.26.0392 Boehringer Ingelheim Investigational Site, Ocean City, New Jersey
  - 1160.26.0472 Boehringer Ingelheim Investigational Site, Paterson, New Jersey
  - 1160.26.0221 Boehringer Ingelheim Investigational Site, Voorhees Township, New Jersey
  - 1160.26.0254 Boehringer Ingelheim Investigational Site, Westwood, New Jersey
  - 1160.26.0127 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1160.26.0423 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1160.26.0476 Boehringer Ingelheim Investigational Site, Albany, New York
  - 1160.26.0063 Boehringer Ingelheim Investigational Site, Buffalo, New York
  - 1160.26.0044 Boehringer Ingelheim Investigational Site, Cortlandt Manor, New York
  - 1160.26.0373 Boehringer Ingelheim Investigational Site, Flushing, New York
  - 1160.26.0045 Boehringer Ingelheim Investigational Site, Garden City, New York
  - 1160.26.0251 Boehringer Ingelheim Investigational Site, Kingston, New York
  - 1160.26.0229 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 1160.26.0451 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 1160.26.0090 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1160.26.0183 Boehringer Ingelheim Investigational Site, New Rochelle, New York
  - 1160.26.0316 Boehringer Ingelheim Investigational Site, New York, New York
  - 1160.26.0146 Boehringer Ingelheim Investigational Site, North Massapequa, New York
  - 1160.26.0210 Boehringer Ingelheim Investigational Site, Northport, New York
  - 1160.26.0075 Boehringer Ingelheim Investigational Site, Poughkeepsie, New York
  - 1160.26.0197 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1160.26.0320 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1160.26.0064 Boehringer Ingelheim Investigational Site, Scarsdale, New York
  - 1160.26.0113 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1160.26.0281 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1160.26.0414 Boehringer Ingelheim Investigational Site, Troy, New York
  - 1160.26.0356 Boehringer Ingelheim Investigational Site, Watertown, New York
  - 1160.26.0039 Boehringer Ingelheim Investigational Site, Williamsville, New York
  - 1160.26.0353 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 1160.26.0080 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1160.26.0412 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1160.26.0350 Boehringer Ingelheim Investigational Site, Gastonia, North Carolina
  - 1160.26.0322 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 1160.26.0173 Boehringer Ingelheim Investigational Site, High Point, North Carolina
  - 1160.26.0108 Boehringer Ingelheim Investigational Site, Lexington, North Carolina
  - 1160.26.0006 Boehringer Ingelheim Investigational Site, Pinehurst, North Carolina
  - 1160.26.0002 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1160.26.0069 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1160.26.0372 Boehringer Ingelheim Investigational Site, Wilmington, North Carolina
  - 1160.26.0094 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1160.26.0425 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1160.26.0102 Boehringer Ingelheim Investigational Site, Grand Forks, North Dakota
  - 1160.26.0222 Boehringer Ingelheim Investigational Site, Jamestown, North Dakota
  - 1160.26.0203 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1160.26.0434 Boehringer Ingelheim Investigational Site, Canal Fulton, Ohio
  - 1160.26.0083 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1160.26.0402 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1160.26.0426 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1160.26.0479 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1160.26.0263 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1160.26.0480 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1160.26.0267 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1160.26.0035 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1160.26.0150 Boehringer Ingelheim Investigational Site, Fairview Park, Ohio
  - 1160.26.0201 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1160.26.0223 Boehringer Ingelheim Investigational Site, Lorain, Ohio
  - 1160.26.0214 Boehringer Ingelheim Investigational Site, Lyndhurst, Ohio
  - 1160.26.0275 Boehringer Ingelheim Investigational Site, Sandusky, Ohio
  - 1160.26.0103 Boehringer Ingelheim Investigational Site, Westlake, Ohio
  - 1160.26.0155 Boehringer Ingelheim Investigational Site, Bartlesville, Oklahoma
  - 1160.26.0435 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1160.26.0139 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1160.26.0325 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1160.26.0078 Boehringer Ingelheim Investigational Site, Hillsboro, Oregon
  - 1160.26.0245 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1160.26.0133 Boehringer Ingelheim Investigational Site, Springfield, Oregon
  - 1160.26.0301 Boehringer Ingelheim Investigational Site, Allentown, Pennsylvania
  - 1160.26.0454 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1160.26.0295 Boehringer Ingelheim Investigational Site, Camp Hill, Pennsylvania
  - 1160.26.0294 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 1160.26.0369 Boehringer Ingelheim Investigational Site, Jenkintown, Pennsylvania
  - 1160.26.0303 Boehringer Ingelheim Investigational Site, Jersey Shore, Pennsylvania
  - 1160.26.0431 Boehringer Ingelheim Investigational Site, Lancaster, Pennsylvania
  - 1160.26.0168 Boehringer Ingelheim Investigational Site, Langhorne, Pennsylvania
  - 1160.26.0293 Boehringer Ingelheim Investigational Site, Meadowbrook, Pennsylvania
  - 1160.26.0025 Boehringer Ingelheim Investigational Site, Newton, Pennsylvania
  - 1160.26.0394 Boehringer Ingelheim Investigational Site, Norristown, Pennsylvania
  - 1160.26.0158 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1160.26.0181 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1160.26.0416 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1160.26.0344 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1160.26.0466 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1160.26.0208 Boehringer Ingelheim Investigational Site, Sellersville, Pennsylvania
  - 1160.26.0465 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1160.26.0400 Boehringer Ingelheim Investigational Site, Upland, Pennsylvania
  - 1160.26.0032 Boehringer Ingelheim Investigational Site, Wynnewood, Pennsylvania
  - 1160.26.0067 Boehringer Ingelheim Investigational Site, Wyomissing, Pennsylvania
  - 1160.26.0212 Boehringer Ingelheim Investigational Site, Pawtucket, Rhode Island
  - 1160.26.0007 Boehringer Ingelheim Investigational Site, Beaufort, South Carolina
  - 1160.26.0383 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1160.26.0313 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1160.26.0450 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 1160.26.0166 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1160.26.0008 Boehringer Ingelheim Investigational Site, Summerville, South Carolina
  - 1160.26.0468 Boehringer Ingelheim Investigational Site, West Columbia, South Carolina
  - 1160.26.0348 Boehringer Ingelheim Investigational Site, Rapid City, South Dakota
  - 1160.26.0084 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1160.26.0062 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 1160.26.0370 Boehringer Ingelheim Investigational Site, Johnson City, Tennessee
  - 1160.26.0323 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1160.26.0395 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1160.26.0474 Boehringer Ingelheim Investigational Site, Oak Ridge, Tennessee
  - 1160.26.0129 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1160.26.0410 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1160.26.0156 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1160.26.0315 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1160.26.0444 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1160.26.0447 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1160.26.0483 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1160.26.0335 Boehringer Ingelheim Investigational Site, Lubbock, Texas
  - 1160.26.0230 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 1160.26.0467 Boehringer Ingelheim Investigational Site, Plano, Texas
  - 1160.26.0013 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1160.26.0269 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1160.26.0307 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1160.26.0285 Boehringer Ingelheim Investigational Site, San Marcos, Texas
  - 1160.26.0215 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 1160.26.0367 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 1160.26.0195 Boehringer Ingelheim Investigational Site, Arlington, Virginia
  - 1160.26.0453 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 1160.26.0053 Boehringer Ingelheim Investigational Site, Chesapeake, Virginia
  - 1160.26.0098 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 1160.26.0386 Boehringer Ingelheim Investigational Site, Falls Church, Virginia
  - 1160.26.0428 Boehringer Ingelheim Investigational Site, Fredericksburg, Virginia
  - 1160.26.0311 Boehringer Ingelheim Investigational Site, Harrisonburg, Virginia
  - 1160.26.0292 Boehringer Ingelheim Investigational Site, Newport News, Virginia
  - 1160.26.0224 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 1160.26.0220 Boehringer Ingelheim Investigational Site, Salem, Virginia
  - 1160.26.0317 Boehringer Ingelheim Investigational Site, Winchester, Virginia
  - 1160.26.0287 Boehringer Ingelheim Investigational Site, Bellevue, Washington
  - 1160.26.0050 Boehringer Ingelheim Investigational Site, Bellingham, Washington
  - 1160.26.0040 Boehringer Ingelheim Investigational Site, Burien, Washington
  - 1160.26.0298 Boehringer Ingelheim Investigational Site, Olympia, Washington
  - 1160.26.0250 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1160.26.0256 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1160.26.0024 Boehringer Ingelheim Investigational Site, Wenatchee, Washington
  - 1160.26.0193 Boehringer Ingelheim Investigational Site, Charleston, West Virginia
  - 1160.26.0169 Boehringer Ingelheim Investigational Site, Clarksburg, West Virginia
  - 1160.26.0365 Boehringer Ingelheim Investigational Site, Huntington, West Virginia
  - 1160.26.0072 Boehringer Ingelheim Investigational Site, Elkhorn, Wisconsin
  - 1160.26.0234 Boehringer Ingelheim Investigational Site, Green Bay, Wisconsin
  - 1160.26.0099 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - 1160.26.0242 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - 1160.26.0359 Boehringer Ingelheim Investigational Site, Marshfield, Wisconsin
  - 1160.26.0461 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Argentina (13):
  - 1160.26.0523 Boehringer Ingelheim Investigational Site, Bahía Blanca
  - 1160.26.0524 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.26.0533 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.26.0526 Boehringer Ingelheim Investigational Site, Cipolletti
  - 1160.26.0529 Boehringer Ingelheim Investigational Site, Coronel Suárez
  - 1160.26.0531 Boehringer Ingelheim Investigational Site, Córdoba
  - 1160.26.0530 Boehringer Ingelheim Investigational Site, La Plata
  - 1160.26.0527 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1160.26.0532 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1160.26.0525 Boehringer Ingelheim Investigational Site, Quilmes
  - 1160.26.0521 Boehringer Ingelheim Investigational Site, Rosario
  - 1160.26.0528 Boehringer Ingelheim Investigational Site, Salta
  - 1160.26.0522 Boehringer Ingelheim Investigational Site, Santa Fe
- Australia (10):
  - 1160.26.0508 Boehringer Ingelheim Investigational Site, Coffs Harbour, New South Wales
  - 1160.26.0510 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 1160.26.0505 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 1160.26.0506 Boehringer Ingelheim Investigational Site, Milton, Queensland
  - 1160.26.0509 Boehringer Ingelheim Investigational Site, Ashford, South Australia
  - 1160.26.0507 Boehringer Ingelheim Investigational Site, Launceston, Tasmania
  - 1160.26.0504 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1160.26.0501 Boehringer Ingelheim Investigational Site, Geelong, Victoria
  - 1160.26.0502 Boehringer Ingelheim Investigational Site, Parkville, Victoria
  - 1160.26.0503 Boehringer Ingelheim Investigational Site, Prahran, Victoria
- Austria (10):
  - 1160.26.0543 Boehringer Ingelheim Investigational Site, Graz
  - 1160.26.0549 Boehringer Ingelheim Investigational Site, Linz
  - 1160.26.0541 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.26.0542 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.26.0544 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.26.0545 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.26.0547 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.26.0548 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.26.0546 Boehringer Ingelheim Investigational Site, Wels
  - 1160.26.0550 Boehringer Ingelheim Investigational Site, Wiener Neustadt
- Belgium (25):
  - 1160.26.0564 Boehringer Ingelheim Investigational Site, Aalst
  - 1160.26.0573 Boehringer Ingelheim Investigational Site, Antwerp
  - 1160.26.0575 Boehringer Ingelheim Investigational Site, Antwerp
  - 1160.26.0572 Boehringer Ingelheim Investigational Site, Brasschaat
  - 1160.26.0577 Boehringer Ingelheim Investigational Site, Bruges
  - 1160.26.0571 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.26.0581 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.26.0585 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.26.0586 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.26.0563 Boehringer Ingelheim Investigational Site, Edegem
  - 1160.26.0578 Boehringer Ingelheim Investigational Site, Genk
  - 1160.26.0587 Boehringer Ingelheim Investigational Site, Genk
  - 1160.26.0574 Boehringer Ingelheim Investigational Site, Ghent
  - 1160.26.0588 Boehringer Ingelheim Investigational Site, Gilly
  - 1160.26.0580 Boehringer Ingelheim Investigational Site, Haine-St.-Paul
  - 1160.26.0568 Boehringer Ingelheim Investigational Site, Hasselt
  - 1160.26.0569 Boehringer Ingelheim Investigational Site, Kortrijk
  - 1160.26.0561 Boehringer Ingelheim Investigational Site, Leuven
  - 1160.26.0579 Boehringer Ingelheim Investigational Site, Liège
  - 1160.26.0583 Boehringer Ingelheim Investigational Site, Liège
  - 1160.26.0589 Boehringer Ingelheim Investigational Site, Mol
  - 1160.26.0567 Boehringer Ingelheim Investigational Site, Ostend
  - 1160.26.0570 Boehringer Ingelheim Investigational Site, Roeselare
  - 1160.26.0566 Boehringer Ingelheim Investigational Site, Tienen
  - 1160.26.0562 Boehringer Ingelheim Investigational Site, Turnhout
- Brazil (14):
  - 1160.26.550648 Boehringer Ingelheim Investigational Site, Belo Horizonte
  - 1160.26.550654 Boehringer Ingelheim Investigational Site, Blumenau
  - 1160.26.550644 Boehringer Ingelheim Investigational Site, Campinas
  - 1160.26.550650 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.26.550651 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.26.550653 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.26.550652 Boehringer Ingelheim Investigational Site, Goiânia
  - 1160.26.550645 Boehringer Ingelheim Investigational Site, Marília
  - 1160.26.550646 Boehringer Ingelheim Investigational Site, São José do Rio Preto
  - 1160.26.550647 Boehringer Ingelheim Investigational Site, São José do Rio Preto
  - 1160.26.550641 Boehringer Ingelheim Investigational Site, São Paulo
  - 1160.26.550642 Boehringer Ingelheim Investigational Site, São Paulo
  - 1160.26.550643 Boehringer Ingelheim Investigational Site, São Paulo
  - 1160.26.550649 Boehringer Ingelheim Investigational Site, Uberaba
- Bulgaria (15):
  - 1160.26.0620 Boehringer Ingelheim Investigational Site, Pleven
  - 1160.26.0611 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0612 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0613 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0614 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0615 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0616 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0617 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0618 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0622 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0623 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0624 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0625 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.26.0626 Boehringer Ingelheim Investigational Site, Stara Zagora
  - 1160.26.0621 Boehringer Ingelheim Investigational Site, Varna
- Canada (54):
  - 1160.26.0694 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1160.26.0696 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1160.26.0680 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1160.26.0712 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1160.26.0706 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 1160.26.0725 Boehringer Ingelheim Investigational Site, Nanaimo, British Columbia
  - 1160.26.0691 Boehringer Ingelheim Investigational Site, New Westminster, British Columbia
  - 1160.26.0714 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1160.26.0701 Boehringer Ingelheim Investigational Site, Portage la Prairie, Manitoba
  - 1160.26.0698 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1160.26.0707 Boehringer Ingelheim Investigational Site, Bay Roberts, Newfoundland and Labrador
  - 1160.26.0676 Boehringer Ingelheim Investigational Site, Antigonish, Nova Scotia
  - 1160.26.0703 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1160.26.0679 Boehringer Ingelheim Investigational Site, Ajax, Ontario
  - 1160.26.0677 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1160.26.0674 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 1160.26.0702 Boehringer Ingelheim Investigational Site, Cambridge, Ontario
  - 1160.26.0720 Boehringer Ingelheim Investigational Site, Cambridge, Ontario
  - 1160.26.0671 Clinical Research & Diagnostic Solutions Inc., Etobicoke, Ontario
  - 1160.26.0715 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1160.26.0692 Boehringer Ingelheim Investigational Site, Grimsby, Ontario
  - 1160.26.0685 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.26.0697 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.26.0710 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.26.0719 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.26.0721 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.26.0689 Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - 1160.26.0695 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1160.26.0708 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1160.26.0724 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1160.26.0688 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1160.26.0672 Boehringer Ingelheim Investigational Site, Oshawa, Ontario
  - 1160.26.0687 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1160.26.0723 Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 1160.26.0690 Boehringer Ingelheim Investigational Site, Thunder Bay, Ontario
  - 1160.26.0684 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.26.0718 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.26.0711 Boehringer Ingelheim Investigational Site, Waterloo, Ontario
  - 1160.26.0686 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 1160.26.0693 Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - 1160.26.0681 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.26.0683 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.26.0705 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.26.0709 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.26.0716 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.26.0717 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1160.26.0713 Boehringer Ingelheim Investigational Site, Saint George-de-Beauce, Quebec
  - 1160.26.0699 Boehringer Ingelheim Investigational Site, Saint-Charles-Borromée, Quebec
  - 1160.26.0675 Boehringer Ingelheim Investigational Site, Saint-Hyacinthe, Quebec
  - 1160.26.0704 Boehringer Ingelheim Investigational Site, Saint-Jérôme, Quebec
  - 1160.26.0700 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
  - 1160.26.0682 Boehringer Ingelheim Investigational Site, Terrebonne (Lachenaie), Quebec
  - 1160.26.0673 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
  - 1160.26.0678 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (13):
  - 1160.26.0771 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.26.0772 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.26.0773 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.26.0774 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.26.0775 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.26.0783 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.26.0784 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1160.26.0776 Boehringer Ingelheim Investigational Site, Harbin
  - 1160.26.0778 Boehringer Ingelheim Investigational Site, Qingdao
  - 1160.26.0781 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.26.0782 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.26.0777 Boehringer Ingelheim Investigational Site, Shenyang
  - 1160.26.0780 Boehringer Ingelheim Investigational Site, Shijiazhuang
- Colombia (3):
  - 1160.26.0801 Boehringer Ingelheim Investigational Site, Bogotá
  - 1160.26.0802 Boehringer Ingelheim Investigational Site, Bogotá
  - 1160.26.0803 Boehringer Ingelheim Investigational Site, Bogotá
- Czechia (10):
  - 1160.26.0815 Boehringer Ingelheim Investigational Site, Brno
  - 1160.26.0816 Boehringer Ingelheim Investigational Site, Brno
  - 1160.26.0820 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.26.0818 Boehringer Ingelheim Investigational Site, Pardubice
  - 1160.26.0814 Boehringer Ingelheim Investigational Site, Plzen-Bory
  - 1160.26.0813 Boehringer Ingelheim Investigational Site, Pragha 9
  - 1160.26.0811 Boehringer Ingelheim Investigational Site, Prague
  - 1160.26.0812 Boehringer Ingelheim Investigational Site, Prague
  - 1160.26.0817 Boehringer Ingelheim Investigational Site, Příbram
  - 1160.26.0819 Boehringer Ingelheim Investigational Site, Ústí nad Orlicí
- Denmark (11):
  - 1160.26.0837 Boehringer Ingelheim Investigational Site, Aalborg
  - 1160.26.0835 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1160.26.0833 Boehringer Ingelheim Investigational Site, Elsinore
  - 1160.26.0838 Boehringer Ingelheim Investigational Site, Frederikssund
  - 1160.26.0834 Boehringer Ingelheim Investigational Site, Herlev
  - 1160.26.0841 Boehringer Ingelheim Investigational Site, Horsens
  - 1160.26.0832 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1160.26.0840 Boehringer Ingelheim Investigational Site, Køge
  - 1160.26.0831 Boehringer Ingelheim Investigational Site, Odense
  - 1160.26.0839 Boehringer Ingelheim Investigational Site, Roskilde
  - 1160.26.0836 Boehringer Ingelheim Investigational Site, Svendborg
- Finland (9):
  - 1160.26.0856 Boehringer Ingelheim Investigational Site, Espoo
  - 1160.26.0851 Boehringer Ingelheim Investigational Site, HUS
  - 1160.26.0859 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1160.26.0855 Boehringer Ingelheim Investigational Site, Kuopio
  - 1160.26.0857 Boehringer Ingelheim Investigational Site, Lappeenranta
  - 1160.26.0854 Boehringer Ingelheim Investigational Site, OYS
  - 1160.26.0858 Boehringer Ingelheim Investigational Site, Pori
  - 1160.26.0852 Boehringer Ingelheim Investigational Site, Tampere
  - 1160.26.0853 Boehringer Ingelheim Investigational Site, Turku
- France (41):
  - 1160.26.0875A Boehringer Ingelheim Investigational Site, Abbeville
  - 1160.26.0882A Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882B Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882C Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882D Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882E Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882G Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882H Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882I Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882K Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0882L Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0884A Boehringer Ingelheim Investigational Site, Angers
  - 1160.26.0887A Boehringer Ingelheim Investigational Site, Cholet
  - 1160.26.0889A Boehringer Ingelheim Investigational Site, Gap
  - 1160.26.0888A Boehringer Ingelheim Investigational Site, Grenoble
  - 1160.26.0880B Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1160.26.0880C Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1160.26.0880D Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1160.26.0880E Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1160.26.0879A Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0879B Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0879C Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0879E Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0879F Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0879G Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0879H Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0879S Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0880A Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0880F Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0880G Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0880J Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0881A Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0881D Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1160.26.0874A Boehringer Ingelheim Investigational Site, Langres
  - 1160.26.0874B Boehringer Ingelheim Investigational Site, Langres
  - 1160.26.0871A Boehringer Ingelheim Investigational Site, Paris
  - 1160.26.0873A Boehringer Ingelheim Investigational Site, Toulouse
  - 1160.26.0886A Boehringer Ingelheim Investigational Site, Tourcoing
  - 1160.26.0872A Boehringer Ingelheim Investigational Site, Valenciennes
  - 1160.26.0872B Boehringer Ingelheim Investigational Site, Valenciennes
  - 1160.26.0872C Boehringer Ingelheim Investigational Site, Valenciennes
- Germany (27):
  - 1160.26.0932 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.26.0948 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.26.0962 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.26.0940 Boehringer Ingelheim Investigational Site, Bochum
  - 1160.26.0936 Boehringer Ingelheim Investigational Site, Coburg
  - 1160.26.0963 Boehringer Ingelheim Investigational Site, Cologne
  - 1160.26.0968 Boehringer Ingelheim Investigational Site, Dachau
  - 1160.26.0972 Boehringer Ingelheim Investigational Site, Dortmund
  - 1160.26.0957 Boehringer Ingelheim Investigational Site, Duisburg
  - 1160.26.0971 Boehringer Ingelheim Investigational Site, Erlangen
  - 1160.26.0965 Boehringer Ingelheim Investigational Site, Eschweiler
  - 1160.26.0934 Boehringer Ingelheim Investigational Site, Essen
  - 1160.26.0931 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1160.26.0943 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1160.26.0955 Boehringer Ingelheim Investigational Site, Kassel
  - 1160.26.0946 Boehringer Ingelheim Investigational Site, Lahr
  - 1160.26.0944 Boehringer Ingelheim Investigational Site, Limburg
  - 1160.26.0951 Boehringer Ingelheim Investigational Site, Mainz
  - 1160.26.0933 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.26.0945 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.26.0970 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.26.0947 Boehringer Ingelheim Investigational Site, München
  - 1160.26.0952 Boehringer Ingelheim Investigational Site, München
  - 1160.26.0941 Boehringer Ingelheim Investigational Site, Papenburg
  - 1160.26.0959 Boehringer Ingelheim Investigational Site, Suhl
  - 1160.26.0937 Boehringer Ingelheim Investigational Site, Witten
  - 1160.26.0966 Boehringer Ingelheim Investigational Site, Wuppertal
- Greece (13):
  - 1160.26.0908 University Hospital of Alexandroupolis, Alexandroupoli
  - 1160.26.0901 General Hospital "Alexandra", Therapeutic Clinic UOA, Athens
  - 1160.26.0906 General Hospital ";Evangelismos", Athens
  - 1160.26.0907 "Pammakaristos" Hospital of Athens, Athens
  - 1160.26.0915 "Hippokratio" Hospital of Athens, Athens
  - 1160.26.0914 2nd IKA Hospital, Thessaloniki, Kalamaria-Thessaloniki
  - 1160.26.0904 General Hospital of Larissa, Larissa
  - 1160.26.0913 University Hospital of Larissa, Larissa
  - 1160.26.0912 General Hospital of Leivadia, Livadeia
  - 1160.26.0910 General Hospital of Thiva, Thebes
  - 1160.26.0902 General Hospital " Papageorgiou", Thessaloniki
  - 1160.26.0903 General Hospital of Trikala, Trikala
  - 1160.26.0905 Boehringer Ingelheim Investigational Site, Voula - Athens
- Hong Kong (4):
  - 1160.26.1001 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1160.26.1002 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1160.26.1003 Boehringer Ingelheim Investigational Site, Kowloon
  - 1160.26.1004 Boehringer Ingelheim Investigational Site, Kowloon
- Hungary (10):
  - 1160.26.1011 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.26.1012 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.26.1013 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.26.1014 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.26.1015 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.26.1016 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.26.1020 Boehringer Ingelheim Investigational Site, Gyöngyös
  - 1160.26.1017 Boehringer Ingelheim Investigational Site, Komárom
  - 1160.26.1018 Boehringer Ingelheim Investigational Site, Pécs
  - 1160.26.1019 Boehringer Ingelheim Investigational Site, Veszprém
- India (20):
  - 1160.26.1056 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1160.26.1057 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1160.26.1064 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.26.1065 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.26.1071 Boehringer Ingelheim Investigational Site, Bikaner
  - 1160.26.1066 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.26.1069 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1160.26.1062 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1160.26.1058 Boehringer Ingelheim Investigational Site, Indore
  - 1160.26.1053 Boehringer Ingelheim Investigational Site, Jaipur
  - 1160.26.1073 Boehringer Ingelheim Investigational Site, Jaipur
  - 1160.26.1067 Boehringer Ingelheim Investigational Site, Kerala
  - 1160.26.1068 Boehringer Ingelheim Investigational Site, Kottayam
  - 1160.26.1055 Boehringer Ingelheim Investigational Site, Lucknow
  - 1160.26.1051 Boehringer Ingelheim Investigational Site, Ludhiana
  - 1160.26.1060 Boehringer Ingelheim Investigational Site, Mumbai
  - 1160.26.1072 Boehringer Ingelheim Investigational Site, Mysore
  - 1160.26.1059 Boehringer Ingelheim Investigational Site, Nagpur
  - 1160.26.1052 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.26.1070 Boehringer Ingelheim Investigational Site, Pune
- Israel (32):
  - 1160.26.1110 Boehringer Ingelheim Investigational Site, Afula
  - 1160.26.1121 Boehringer Ingelheim Investigational Site, Afula
  - 1160.26.1111 Boehringer Ingelheim Investigational Site, Ashkelon
  - 1160.26.1102 Boehringer Ingelheim Investigational Site, Beersheba
  - 1160.26.1117 Boehringer Ingelheim Investigational Site, Giv‘atayim
  - 1160.26.1112 Boehringer Ingelheim Investigational Site, Hadera
  - 1160.26.1091 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.26.1113 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.26.1114 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.26.1116 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.26.1118 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.26.1105 Boehringer Ingelheim Investigational Site, Holon
  - 1160.26.1097 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1160.26.1101 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1160.26.1104 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1160.26.1106 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1160.26.1119 Boehringer Ingelheim Investigational Site, Kfar Saba
  - 1160.26.1115 Boehringer Ingelheim Investigational Site, Nazareth
  - 1160.26.1096 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1160.26.1093 Boehringer Ingelheim Investigational Site, Ramat Gan
  - 1160.26.1094 Boehringer Ingelheim Investigational Site, Ramat Gan
  - 1160.26.1095 Boehringer Ingelheim Investigational Site, Ramat Gan
  - 1160.26.1100 Boehringer Ingelheim Investigational Site, Rehovot
  - 1160.26.1103 Boehringer Ingelheim Investigational Site, Safed
  - 1160.26.1107 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.26.1108 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.26.1109 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.26.1120 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.26.1122 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.26.1092 Boehringer Ingelheim Investigational Site, Tel Litwinsky
  - 1160.26.1098 Boehringer Ingelheim Investigational Site, Tel Litwinsky
  - 1160.26.1099 Boehringer Ingelheim Investigational Site, Ẕerifin
- Italy (18):
  - 1160.26.1169 Boehringer Ingelheim Investigational Site, Arezzo
  - 1160.26.1172 Boehringer Ingelheim Investigational Site, Ascoli Piceno
  - 1160.26.1180 Boehringer Ingelheim Investigational Site, Bentivoglio (BO)
  - 1160.26.1161 Boehringer Ingelheim Investigational Site, Bologna
  - 1160.26.1163 Boehringer Ingelheim Investigational Site, Castelnuovo Garfagnana
  - 1160.26.1178 Boehringer Ingelheim Investigational Site, Chieti
  - 1160.26.1171 Boehringer Ingelheim Investigational Site, Colleferro
  - 1160.26.1174 Boehringer Ingelheim Investigational Site, Cremona
  - 1160.26.1167 Boehringer Ingelheim Investigational Site, Eboli
  - 1160.26.1168 Boehringer Ingelheim Investigational Site, Isernia
  - 1160.26.1162 Boehringer Ingelheim Investigational Site, Legnago
  - 1160.26.1177 Boehringer Ingelheim Investigational Site, Mantova
  - 1160.26.1165 Boehringer Ingelheim Investigational Site, Perugia SAN Sisto
  - 1160.26.1175 Boehringer Ingelheim Investigational Site, Roma
  - 1160.26.1181 Boehringer Ingelheim Investigational Site, San Bonifacio
  - 1160.26.1173 Boehringer Ingelheim Investigational Site, San Daniele del Friuli
  - 1160.26.1170 Boehringer Ingelheim Investigational Site, Sassari
  - 1160.26.1176 Boehringer Ingelheim Investigational Site, Sassari
- Japan (49):
  - 1160.26.1204 Boehringer Ingelheim Investigational Site, Abeno-ku, Osaka, Osaka
  - 1160.26.1209 Boehringer Ingelheim Investigational Site, Aki-gun, Hiroshima
  - 1160.26.1193 Boehringer Ingelheim Investigational Site, Aoba-ku, Sendai, Miyagi
  - 1160.26.1211 Boehringer Ingelheim Investigational Site, Chuo-ku, Fukuoka, Fukuoka
  - 1160.26.1225 Boehringer Ingelheim Investigational Site, Chuo-ku, Fukuoka, Fukuoka
  - 1160.26.1221 Boehringer Ingelheim Investigational Site, Chuo-ku, Kobe, Hyogo
  - 1160.26.1219 Boehringer Ingelheim Investigational Site, Chuo-ku, Osaka, Osaka
  - 1160.26.1229 Boehringer Ingelheim Investigational Site, Fujioka-shi , Gunma-ken
  - 1160.26.1232 Boehringer Ingelheim Investigational Site, Fukushima-shi,Fukushima-ken
  - 1160.26.1228 Boehringer Ingelheim Investigational Site, Higashimatsushimashi, Miyagi-ken
  - 1160.26.1208 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1160.26.1214 Boehringer Ingelheim Investigational Site, Iida, Nagano
  - 1160.26.1240 Boehringer Ingelheim Investigational Site, Isesaki-shi,Gunma
  - 1160.26.1224 Boehringer Ingelheim Investigational Site, Iwakuni, Yamaguchi
  - 1160.26.1194 Boehringer Ingelheim Investigational Site, Izumi-ku, Sendai, Miyagi
  - 1160.26.1241 Boehringer Ingelheim Investigational Site, Kamigyo-ku, Kyoto
  - 1160.26.1220 Boehringer Ingelheim Investigational Site, Kawachinagano, Osaka
  - 1160.26.1203 Boehringer Ingelheim Investigational Site, Kita-ku, Osaka, Osaka
  - 1160.26.1207 Boehringer Ingelheim Investigational Site, Kita-ku, Sakai, Osaka
  - 1160.26.1231 Boehringer Ingelheim Investigational Site, Komatsu-shi,Ishikawa -ken
  - 1160.26.1233 Boehringer Ingelheim Investigational Site, Kyoto-shi,Kyoto
  - 1160.26.1242 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1160.26.1210 Boehringer Ingelheim Investigational Site, Minami-ku, Fukuoka, Fukuoka
  - 1160.26.1218 Boehringer Ingelheim Investigational Site, Minato, Tokyo
  - 1160.26.1200 Boehringer Ingelheim Investigational Site, Minato-ku, Nagoya, Aichi
  - 1160.26.1201 Boehringer Ingelheim Investigational Site, Minato-ku, Nagoya, Aichi
  - 1160.26.1216 Boehringer Ingelheim Investigational Site, Narashino, Chiba
  - 1160.26.1237 Boehringer Ingelheim Investigational Site, Nishinomiya-shi,Hyogo
  - 1160.26.1223 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 1160.26.1197 Boehringer Ingelheim Investigational Site, Oota, Tokyo
  - 1160.26.1212 Boehringer Ingelheim Investigational Site, Otaru, Hokkaido
  - 1160.26.1230 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa-ken
  - 1160.26.1238 Boehringer Ingelheim Investigational Site, Sapporo-shi,Hokkai-do
  - 1160.26.1217 Boehringer Ingelheim Investigational Site, Shibuya, Tokyo
  - 1160.26.1196 Boehringer Ingelheim Investigational Site, Shinjuku, Tokyo
  - 1160.26.1191 Boehringer Ingelheim Investigational Site, Shiroishi-ku, Sapporo, Hokkaido
  - 1160.26.1192 Boehringer Ingelheim Investigational Site, Shiroishi-ku, Sapporo, Hokkaido
  - 1160.26.1206 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1160.26.1235 Boehringer Ingelheim Investigational Site, Suita-shi, Osaka
  - 1160.26.1236 Boehringer Ingelheim Investigational Site, Suita-shi, Osaka
  - 1160.26.1205 Boehringer Ingelheim Investigational Site, Sumiyoshi-ku, Osaka, Osaka
  - 1160.26.1234 Boehringer Ingelheim Investigational Site, Takatsuki-shi,Osaka
  - 1160.26.1215 Boehringer Ingelheim Investigational Site, Tokorozawa, Saitama
  - 1160.26.1198 Boehringer Ingelheim Investigational Site, Totsuka-ku, Yokohama, Kanagawa
  - 1160.26.1195 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaragi
  - 1160.26.1199 Boehringer Ingelheim Investigational Site, Ueda, Nagano
  - 1160.26.1222 Boehringer Ingelheim Investigational Site, Wakayama, Wakayama
  - 1160.26.1227 Boehringer Ingelheim Investigational Site, Yanagawa, Fukuoka
  - 1160.26.1243 Boehringer Ingelheim Investigational Site, Yao, Osaka
- Malaysia (7):
  - 1160.26.1295 Boehringer Ingelheim Investigational Site, George Town
  - 1160.26.1296 Boehringer Ingelheim Investigational Site, George Town
  - 1160.26.1297 Boehringer Ingelheim Investigational Site, Kajang,Selangor
  - 1160.26.1291 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1160.26.1292 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1160.26.1294 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1160.26.1293 Boehringer Ingelheim Investigational Site, Kuching
- Mexico (8):
  - 1160.26.1318 Hospital General "Dr. Santiago Ramón y Cajal, Durango
  - 1160.26.1311 Hospital Mexico-Americano, Guadalajara
  - 1160.26.1317 hOSPITAL bERNARDETTE, Guadalajara
  - 1160.26.1312 Hospital de Jesus, México
  - 1160.26.1314 Hospital 1o. de Octubre, México
  - 1160.26.1319 Instituto Nacional de Cardiologia, México
  - 1160.26.1313 Hosp. Angeles Centro Medico del Potosi, San Luis Potosí City
  - 1160.26.1322 Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
- Netherlands (31):
  - 1160.26.1337 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1160.26.1344 Boehringer Ingelheim Investigational Site, Almelo
  - 1160.26.1331 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.26.1336 Boehringer Ingelheim Investigational Site, Apeldoorn
  - 1160.26.1332 Boehringer Ingelheim Investigational Site, Breda
  - 1160.26.1349 Boehringer Ingelheim Investigational Site, Den Helder
  - 1160.26.1345 Boehringer Ingelheim Investigational Site, Deventer
  - 1160.26.1360 Boehringer Ingelheim Investigational Site, Dirksland
  - 1160.26.1348 Boehringer Ingelheim Investigational Site, Dordrecht
  - 1160.26.1340 Boehringer Ingelheim Investigational Site, Ede
  - 1160.26.1358 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1160.26.1338 Boehringer Ingelheim Investigational Site, Enschede
  - 1160.26.1343 Boehringer Ingelheim Investigational Site, Goes
  - 1160.26.1347 Boehringer Ingelheim Investigational Site, Gorinchem
  - 1160.26.1333 Boehringer Ingelheim Investigational Site, Groningen
  - 1160.26.1355 Boehringer Ingelheim Investigational Site, Groningen
  - 1160.26.1361 Boehringer Ingelheim Investigational Site, Heerlen
  - 1160.26.1339 Boehringer Ingelheim Investigational Site, Hengelo
  - 1160.26.1346 Boehringer Ingelheim Investigational Site, Hilversum
  - 1160.26.1356 Boehringer Ingelheim Investigational Site, Hoorn
  - 1160.26.1359 Boehringer Ingelheim Investigational Site, Maastricht
  - 1160.26.1341 Boehringer Ingelheim Investigational Site, Meppel
  - 1160.26.1354 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1160.26.1351 Boehringer Ingelheim Investigational Site, Sneek
  - 1160.26.1334 Boehringer Ingelheim Investigational Site, Spiijkenisse
  - 1160.26.1335 Boehringer Ingelheim Investigational Site, Terneuzen
  - 1160.26.1353 Boehringer Ingelheim Investigational Site, Tiel
  - 1160.26.1352 Boehringer Ingelheim Investigational Site, Tilburg
  - 1160.26.1350 Boehringer Ingelheim Investigational Site, Veldhoven
  - 1160.26.1342 Boehringer Ingelheim Investigational Site, Velp
  - 1160.26.1357 Boehringer Ingelheim Investigational Site, Venlo
- Norway (7):
  - 1160.26.1396 Boehringer Ingelheim Investigational Site, Gjøvik
  - 1160.26.1393 Boehringer Ingelheim Investigational Site, Moss
  - 1160.26.1395 Boehringer Ingelheim Investigational Site, Nordbyhagen
  - 1160.26.1391 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.26.1392 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.26.1397 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.26.1394 Boehringer Ingelheim Investigational Site, Rud
- Peru (5):
  - 1160.26.1415 Hospital Alberto Sabogal, Bella Vista
  - 1160.26.1411 Clinica San Felipe, Jesús María
  - 1160.26.1412 Clínica Anglo Americana, San Isidro
  - 1160.26.1413 Hospital Cayetano Heredia, San Martín de Porres
  - 1160.26.1414 Clínica Vesalio, Urbanización Sto Tomas de San Borja
- Philippines (5):
  - 1160.26.1421 Philippine General Hospital, Manila
  - 1160.26.1422 Manila Doctors Hospital, Manila
  - 1160.26.1424 The Medical City, Pasig
  - 1160.26.1423 Philippine Heart Center, Quezon City
  - 1160.26.1425 St Lukes Medical Center, Quezon City
- Poland (10):
  - 1160.26.1436 Boehringer Ingelheim Investigational Site, Gdynia
  - 1160.26.1438 Boehringer Ingelheim Investigational Site, Gdynia
  - 1160.26.1437 Boehringer Ingelheim Investigational Site, Gdynia Redlowo
  - 1160.26.1435 Boehringer Ingelheim Investigational Site, Katowice
  - 1160.26.1439 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.26.1440 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.26.1433 Boehringer Ingelheim Investigational Site, Puławy
  - 1160.26.1431 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.26.1432 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.26.1434 Boehringer Ingelheim Investigational Site, Zabrze
- Portugal (9):
  - 1160.26.1456 Boehringer Ingelheim Investigational Site, Amadora
  - 1160.26.1451 Boehringer Ingelheim Investigational Site, Carnaxide
  - 1160.26.1454 Boehringer Ingelheim Investigational Site, Coimbra
  - 1160.26.1459 Boehringer Ingelheim Investigational Site, Coimbra
  - 1160.26.1457 Boehringer Ingelheim Investigational Site, Covilha
  - 1160.26.1453 Boehringer Ingelheim Investigational Site, Lisbon
  - 1160.26.1458 Boehringer Ingelheim Investigational Site, Lisbon
  - 1160.26.1455 Boehringer Ingelheim Investigational Site, Porto
  - 1160.26.1452 Boehringer Ingelheim Investigational Site, Setúbal
- Romania (3):
  - 1160.26.1471 Boehringer Ingelheim Investigational Site, Bucharest
  - 1160.26.1472 Boehringer Ingelheim Investigational Site, Bucharest
  - 1160.26.1478 Boehringer Ingelheim Investigational Site, Cluj-Napoca
- Russia (15):
  - 1160.26.1501 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1502 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1503 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1504 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1505 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1506 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1507 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1508 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1509 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1510 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1511 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.26.1512 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.26.1513 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.26.1514 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.26.1515 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Singapore (2):
  - 1160.26.1531 Boehringer Ingelheim Investigational Site, Singapore
  - 1160.26.1532 Boehringer Ingelheim Investigational Site, Singapore
- Slovakia (10):
  - 1160.26.1548 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1160.26.1541 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.26.1542 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.26.1543 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.26.1544 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.26.1545 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.26.1546 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.26.1549 Boehringer Ingelheim Investigational Site, Košice
  - 1160.26.1550 Boehringer Ingelheim Investigational Site, Košice
  - 1160.26.1547 Boehringer Ingelheim Investigational Site, Žilina
- South Africa (9):
  - 1160.26.1562 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 1160.26.1569 Boehringer Ingelheim Investigational Site, Boksburg
  - 1160.26.1561 Boehringer Ingelheim Investigational Site, Cape Town
  - 1160.26.1564 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.26.1567 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.26.1568 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.26.1566 Boehringer Ingelheim Investigational Site, Pretoria
  - 1160.26.1563 Boehringer Ingelheim Investigational Site, Randburg
  - 1160.26.1565 Boehringer Ingelheim Investigational Site, Somerset West
- South Korea (12):
  - 1160.26.1585 Boehringer Ingelheim Investigational Site, Busan
  - 1160.26.1586 Boehringer Ingelheim Investigational Site, Chungchungnam-Do
  - 1160.26.1584 Boehringer Ingelheim Investigational Site, Daegu
  - 1160.26.1591 Boehringer Ingelheim Investigational Site, Daegu
  - 1160.26.1590 Boehringer Ingelheim Investigational Site, Gwangju
  - 1160.26.1581 Boehringer Ingelheim Investigational Site, Incheon
  - 1160.26.1582 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.26.1583 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.26.1588 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.26.1589 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.26.1592 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.26.1593 Boehringer Ingelheim Investigational Site, Seoul
- Spain (9):
  - 1160.26.1601 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.26.1606 Boehringer Ingelheim Investigational Site, Cadiz
  - 1160.26.1607 Boehringer Ingelheim Investigational Site, Fuenlabrada (Madrid)
  - 1160.26.1604 Boehringer Ingelheim Investigational Site, Leganés, Madrid
  - 1160.26.1603 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.26.1608 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.26.1609 Boehringer Ingelheim Investigational Site, Madrid-San Lorenzo Del Escorial
  - 1160.26.1605 Boehringer Ingelheim Investigational Site, Móstoles (Madrid)
  - 1160.26.1602 Boehringer Ingelheim Investigational Site, Sabadell
- Sweden (14):
  - 1160.26.1633 Sahlgrenska Sjukhuset, Göteboerg
  - 1160.26.1629 AVK-mott, Spec.M1, Länssjukhuset Ryhov, Jönköping
  - 1160.26.1631 Universitetssjukhuset i Linköping, Linköping
  - 1160.26.1627 Hjärtmott. ING 35, Malmö Universitetssjukhus MAS, Malmo
  - 1160.26.1628 Rådhusg. 29, Lars Mörlids Läkarmottagning, Nässjö
  - 1160.26.1625 Hjärtmott./Medicinkliniken, Vrinnevisjukhuset, Norrköping
  - 1160.26.1623 Kardiologiska kliniken, Universitetssjukhuset, Örebro
  - 1160.26.1626 Hjärtkärllaboratoriet, Danderyds Sjukhus AB, Stockholm
  - 1160.26.1632 Capio S:t Görans Sjukhus, Stockholm
  - 1160.26.1634 Södersjukhuset, Stockholm
  - 1160.26.1624 Klin. forskningscentrum, Norrlands Universitetssjukhus, Umeå
  - 1160.26.1621 Kardiologiska kliniken, Akademiska Sjukhuset, Uppsala
  - 1160.26.1635 UCR/Uppsala, Uppsala
  - 1160.26.1622 Hjärtmottagningen, Centrallasarettet, Västerås
- Switzerland (4):
  - 1160.26.1652 Boehringer Ingelheim Investigational Site, Basel
  - 1160.26.1655 Boehringer Ingelheim Investigational Site, Bellinzona
  - 1160.26.1651 Boehringer Ingelheim Investigational Site, Bern
  - 1160.26.1654 Boehringer Ingelheim Investigational Site, Lugano
- Taiwan (13):
  - 1160.26.1680 Boehringer Ingelheim Investigational Site, Changhua County
  - 1160.26.1683 Boehringer Ingelheim Investigational Site, Hualien City
  - 1160.26.1682 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1160.26.1679 China Medical University Hospital, Taichung
  - 1160.26.1681 Boehringer Ingelheim Investigational Site, Tainan
  - 1160.26.1671 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.26.1672 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.26.1673 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.26.1674 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.26.1675 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.26.1676 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.26.1677 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.26.1678 Boehringer Ingelheim Investigational Site, Taoyuan District
- Thailand (5):
  - 1160.26.1701 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.26.1702 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.26.1703 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 1160.26.1704 Boehringer Ingelheim Investigational Site, Khon Kaen
  - 1160.26.1705 Boehringer Ingelheim Investigational Site, Muang Nakhonratchasima
- Turkey (Türkiye) (4):
  - 1160.26.1715 Boehringer Ingelheim Investigational Site, Adana
  - 1160.26.1711 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.26.1713 Gazi Universitesi Tip Fakultesi Kardiyoloji Abd, Ankara
  - 1160.26.1714 Dokuz Eylul Universitesi Tip Fakultesi, Izmir
- Ukraine (11):
  - 1160.26.1727 Boehringer Ingelheim Investigational Site, Dnyepropetrovsk
  - 1160.26.1724 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1160.26.1725 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1160.26.1726 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1160.26.1721 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.26.1722 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.26.1723 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.26.1728 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.26.1730 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.26.1731 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.26.1729 Boehringer Ingelheim Investigational Site, Lviv
- United Kingdom (16):
  - 1160.26.1744 Boehringer Ingelheim Investigational Site, Birmingham
  - 1160.26.1746 Boehringer Ingelheim Investigational Site, Chertsey
  - 1160.26.1747 Boehringer Ingelheim Investigational Site, Glasgow
  - 1160.26.1750 Boehringer Ingelheim Investigational Site, Harrow
  - 1160.26.1753 Boehringer Ingelheim Investigational Site, Hull
  - 1160.26.1755 Boehringer Ingelheim Investigational Site, Kirkcaldy, Fife
  - 1160.26.1741 Boehringer Ingelheim Investigational Site, London
  - 1160.26.1756 Boehringer Ingelheim Investigational Site, London
  - 1160.26.1749 Boehringer Ingelheim Investigational Site, Londonderry
  - 1160.26.1742 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1160.26.1751 Boehringer Ingelheim Investigational Site, Newport
  - 1160.26.1752 Boehringer Ingelheim Investigational Site, Northampton
  - 1160.26.1745 Boehringer Ingelheim Investigational Site, Portadown, County Atrim
  - 1160.26.1743 Boehringer Ingelheim Investigational Site, Romford, Essex
  - 1160.26.1754 Boehringer Ingelheim Investigational Site, Stoke-on-Trent
  - 1160.26.1748 Boehringer Ingelheim Investigational Site, York

REFERENCES:
- [Derived] Hijazi Z, Lindback J, Oldgren J, Benz AP, Alexander JH, Connolly SJ, Eikelboom JW, Granger CB, Lopes RD, Siegbahn A, Wallentin L. Individual net clinical outcome with oral anticoagulation in atrial fibrillation using the ABC-AF risk scores. Am Heart J. 2023 Jul;261:55-63. doi: 10.1016/j.ahj.2023.03.012. Epub 2023 Mar 27. PMID 36990261
- [Derived] Reinhardt SW, Desai NR, Tang Y, Jones PG, Ader J, Spertus JA. Personalizing the decision of dabigatran versus warfarin in atrial fibrillation: A secondary analysis of the Randomized Evaluation of Long-term anticoagulation therapY (RE-LY) trial. PLoS One. 2021 Aug 19;16(8):e0256338. doi: 10.1371/journal.pone.0256338. eCollection 2021. PMID 34411158
- [Derived] Pol T, Hijazi Z, Lindback J, Oldgren J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Granger CB, Lopes RD, Yusuf S, Siegbahn A, Wallentin L. Using multimarker screening to identify biomarkers associated with cardiovascular death in patients with atrial fibrillation. Cardiovasc Res. 2022 Jul 20;118(9):2112-2123. doi: 10.1093/cvr/cvab262. PMID 34358298
- [Derived] Millenaar D, Schumacher H, Brueckmann M, Eikelboom JW, Ezekowitz M, Slawik J, Ewen S, Ukena C, Wallentin L, Connolly S, Yusuf S, Bohm M. Cardiovascular Outcomes According to Polypharmacy and Drug Adherence in Patients with Atrial Fibrillation on Long-Term Anticoagulation (from the RE-LY Trial). Am J Cardiol. 2021 Jun 15;149:27-35. doi: 10.1016/j.amjcard.2021.03.024. Epub 2021 Mar 20. PMID 33757788
- [Derived] Pol T, Hijazi Z, Lindback J, Alexander JH, Bahit MC, De Caterina R, Eikelboom JW, Ezekowitz MD, Gersh BJ, Granger CB, Hylek EM, Lopes R, Siegbahn A, Wallentin L. Evaluation of the prognostic value of GDF-15, ABC-AF-bleeding score and ABC-AF-death score in patients with atrial fibrillation across different geographical areas. Open Heart. 2021 Mar;8(1):e001471. doi: 10.1136/openhrt-2020-001471. PMID 33741689
- [Derived] Hijazi Z, Wallentin L, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Granger CB, Lopes RD, Pol T, Yusuf S, Oldgren J, Siegbahn A. Screening of Multiple Biomarkers Associated With Ischemic Stroke in Atrial Fibrillation. J Am Heart Assoc. 2020 Dec 15;9(24):e018984. doi: 10.1161/JAHA.120.018984. Epub 2020 Dec 9. PMID 33292046
- [Derived] Wallentin L, Lindback J, Eriksson N, Hijazi Z, Eikelboom JW, Ezekowitz MD, Granger CB, Lopes RD, Yusuf S, Oldgren J, Siegbahn A. Angiotensin-converting enzyme 2 (ACE2) levels in relation to risk factors for COVID-19 in two large cohorts of patients with atrial fibrillation. Eur Heart J. 2020 Nov 1;41(41):4037-4046. doi: 10.1093/eurheartj/ehaa697. PMID 32984892
- [Derived] Bohm M, Brueckmann M, Eikelboom JW, Ezekowitz M, Frassdorf M, Hijazi Z, Hohnloser SH, Mahfoud F, Schmieder RE, Schumacher H, Wallentin L, Yusuf S. Cardiovascular outcomes, bleeding risk, and achieved blood pressure in patients on long-term anticoagulation with the thrombin antagonist dabigatran or warfarin: data from the RE-LY trial. Eur Heart J. 2020 Aug 7;41(30):2848-2859. doi: 10.1093/eurheartj/ehaa247. PMID 32385506
- [Derived] Stam-Slob MC, Connolly SJ, van der Graaf Y, van der Leeuw J, Dorresteijn JAN, Eikelboom JW, Peters RJG, Alings M, Visseren FLJ. Individual Treatment Effect Estimation of 2 Doses of Dabigatran on Stroke and Major Bleeding in Atrial Fibrillation. Circulation. 2019 Jun 18;139(25):2846-2856. doi: 10.1161/CIRCULATIONAHA.118.035266. Epub 2019 May 3. PMID 31046423
- [Derived] Hijazi Z, Verdecchia P, Oldgren J, Andersson U, Reboldi G, Di Pasquale G, Mazzotta G, Angeli F, Eikelboom JW, Ezekowitz MD, Connolly SJ, Yusuf S, Wallentin L. Cardiac Biomarkers and Left Ventricular Hypertrophy in Relation to Outcomes in Patients With Atrial Fibrillation: Experiences From the RE - LY Trial. J Am Heart Assoc. 2019 Jan 22;8(2):e010107. doi: 10.1161/JAHA.118.010107. PMID 30651032
- [Derived] Kent AP, Brueckmann M, Fraessdorf M, Connolly SJ, Yusuf S, Eikelboom JW, Oldgren J, Reilly PA, Wallentin L, Ezekowitz MD. Concomitant Oral Anticoagulant and Nonsteroidal Anti-Inflammatory Drug Therapy in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2018 Jul 17;72(3):255-267. doi: 10.1016/j.jacc.2018.04.063. Epub 2018 Jul 9. PMID 30012318
- [Derived] Hijazi Z, Hohnloser SH, Oldgren J, Andersson U, Connolly SJ, Eikelboom JW, Ezekowitz MD, Reilly PA, Yusuf S, Wallentin L. Efficacy and safety of dabigatran compared with warfarin in patients with atrial fibrillation in relation to renal function over time-A RE-LY trial analysis. Am Heart J. 2018 Apr;198:169-177. doi: 10.1016/j.ahj.2017.10.015. Epub 2018 Jan 5. No abstract available. PMID 29653640
- [Derived] Hijazi Z, Oldgren J, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Held C, Hylek EM, Lopes RD, Yusuf S, Granger CB, Siegbahn A, Wallentin L; ARISTOTLE and RE-LY Investigators. A biomarker-based risk score to predict death in patients with atrial fibrillation: the ABC (age, biomarkers, clinical history) death risk score. Eur Heart J. 2018 Feb 7;39(6):477-485. doi: 10.1093/eurheartj/ehx584. PMID 29069359
- [Derived] Verdecchia P, Reboldi G, Angeli F, Mazzotta G, Lip GYH, Brueckmann M, Kleine E, Wallentin L, Ezekowitz MD, Yusuf S, Connolly SJ, Di Pasquale G. Dabigatran vs. warfarin in relation to the presence of left ventricular hypertrophy in patients with atrial fibrillation- the Randomized Evaluation of Long-term anticoagulation therapY (RE-LY) study. Europace. 2018 Feb 1;20(2):253-262. doi: 10.1093/europace/eux022. PMID 28520924
- [Derived] Lauw MN, Eikelboom JW, Coppens M, Wallentin L, Yusuf S, Ezekowitz M, Oldgren J, Nakamya J, Wang J, Connolly SJ. Effects of dabigatran according to age in atrial fibrillation. Heart. 2017 Jul;103(13):1015-1023. doi: 10.1136/heartjnl-2016-310358. Epub 2017 Feb 17. PMID 28213368
- [Derived] Oldgren J, Hijazi Z, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Granger CB, Hylek EM, Lopes RD, Siegbahn A, Yusuf S, Wallentin L; RE-LY and ARISTOTLE Investigators. Performance and Validation of a Novel Biomarker-Based Stroke Risk Score for Atrial Fibrillation. Circulation. 2016 Nov 29;134(22):1697-1707. doi: 10.1161/CIRCULATIONAHA.116.022802. Epub 2016 Aug 28. PMID 27569438
- [Derived] Ezekowitz MD, Nagarakanti R, Noack H, Brueckmann M, Litherland C, Jacobs M, Clemens A, Reilly PA, Connolly SJ, Yusuf S, Wallentin L. Comparison of Dabigatran and Warfarin in Patients With Atrial Fibrillation and Valvular Heart Disease: The RE-LY Trial (Randomized Evaluation of Long-Term Anticoagulant Therapy). Circulation. 2016 Aug 23;134(8):589-98. doi: 10.1161/CIRCULATIONAHA.115.020950. Epub 2016 Aug 5. PMID 27496855
- [Derived] Hijazi Z, Oldgren J, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Held C, Hylek EM, Lopes RD, Siegbahn A, Yusuf S, Granger CB, Wallentin L; ARISTOTLE and RE-LY Investigators. The novel biomarker-based ABC (age, biomarkers, clinical history)-bleeding risk score for patients with atrial fibrillation: a derivation and validation study. Lancet. 2016 Jun 4;387(10035):2302-2311. doi: 10.1016/S0140-6736(16)00741-8. Epub 2016 Apr 4. PMID 27056738
- [Derived] Siegbahn A, Oldgren J, Andersson U, Ezekowitz MD, Reilly PA, Connolly SJ, Yusuf S, Wallentin L, Eikelboom JW. D-dimer and factor VIIa in atrial fibrillation - prognostic values for cardiovascular events and effects of anticoagulation therapy. A RE-LY substudy. Thromb Haemost. 2016 May 2;115(5):921-30. doi: 10.1160/TH15-07-0529. Epub 2016 Jan 28. PMID 26818781
- [Derived] Aulin J, Siegbahn A, Hijazi Z, Ezekowitz MD, Andersson U, Connolly SJ, Huber K, Reilly PA, Wallentin L, Oldgren J. Interleukin-6 and C-reactive protein and risk for death and cardiovascular events in patients with atrial fibrillation. Am Heart J. 2015 Dec;170(6):1151-60. doi: 10.1016/j.ahj.2015.09.018. Epub 2015 Oct 3. PMID 26678637
- [Derived] Brambatti M, Darius H, Oldgren J, Clemens A, Noack HH, Brueckmann M, Yusuf S, Wallentin L, Ezekowitz MD, Connolly SJ, Healey JS. Comparison of dabigatran versus warfarin in diabetic patients with atrial fibrillation: Results from the RE-LY trial. Int J Cardiol. 2015 Oct 1;196:127-31. doi: 10.1016/j.ijcard.2015.05.141. Epub 2015 May 28. PMID 26093161
- [Derived] Bohm M, Ezekowitz MD, Connolly SJ, Eikelboom JW, Hohnloser SH, Reilly PA, Schumacher H, Brueckmann M, Schirmer SH, Kratz MT, Yusuf S, Diener HC, Hijazi Z, Wallentin L. Changes in Renal Function in Patients With Atrial Fibrillation: An Analysis From the RE-LY Trial. J Am Coll Cardiol. 2015 Jun 16;65(23):2481-93. doi: 10.1016/j.jacc.2015.03.577. PMID 26065986
- [Derived] Hijazi Z, Oldgren J, Andersson U, Connolly SJ, Ezekowitz MD, Hohnloser SH, Reilly PA, Siegbahn A, Yusuf S, Wallentin L. Importance of persistent elevation of cardiac biomarkers in atrial fibrillation: a RE-LY substudy. Heart. 2014 Aug;100(15):1193-200. doi: 10.1136/heartjnl-2013-304872. Epub 2014 May 2. PMID 24794140
- [Derived] Verdecchia P, Reboldi G, Di Pasquale G, Mazzotta G, Ambrosio G, Yang S, Pogue J, Wallentin L, Ezekowitz MD, Connolly SJ, Yusuf S; RE-LY Study Investigators. Prognostic usefulness of left ventricular hypertrophy by electrocardiography in patients with atrial fibrillation (from the Randomized Evaluation of Long-Term Anticoagulant Therapy Study). Am J Cardiol. 2014 Feb 15;113(4):669-75. doi: 10.1016/j.amjcard.2013.10.045. Epub 2013 Nov 23. PMID 24359765
- [Derived] Hijazi Z, Hohnloser SH, Oldgren J, Andersson U, Connolly SJ, Eikelboom JW, Ezekowitz MD, Reilly PA, Siegbahn A, Yusuf S, Wallentin L. Efficacy and safety of dabigatran compared with warfarin in relation to baseline renal function in patients with atrial fibrillation: a RE-LY (Randomized Evaluation of Long-term Anticoagulation Therapy) trial analysis. Circulation. 2014 Mar 4;129(9):961-70. doi: 10.1161/CIRCULATIONAHA.113.003628. Epub 2013 Dec 9. PMID 24323795
- [Derived] Majeed A, Hwang HG, Connolly SJ, Eikelboom JW, Ezekowitz MD, Wallentin L, Brueckmann M, Fraessdorf M, Yusuf S, Schulman S. Management and outcomes of major bleeding during treatment with dabigatran or warfarin. Circulation. 2013 Nov 19;128(21):2325-32. doi: 10.1161/CIRCULATIONAHA.113.002332. Epub 2013 Sep 30. PMID 24081972
- [Derived] Reilly PA, Lehr T, Haertter S, Connolly SJ, Yusuf S, Eikelboom JW, Ezekowitz MD, Nehmiz G, Wang S, Wallentin L; RE-LY Investigators. The effect of dabigatran plasma concentrations and patient characteristics on the frequency of ischemic stroke and major bleeding in atrial fibrillation patients: the RE-LY Trial (Randomized Evaluation of Long-Term Anticoagulation Therapy). J Am Coll Cardiol. 2014 Feb 4;63(4):321-8. doi: 10.1016/j.jacc.2013.07.104. Epub 2013 Sep 27. PMID 24076487
- [Derived] Marijon E, Le Heuzey JY, Connolly S, Yang S, Pogue J, Brueckmann M, Eikelboom J, Themeles E, Ezekowitz M, Wallentin L, Yusuf S; RE-LY Investigators. Causes of death and influencing factors in patients with atrial fibrillation: a competing-risk analysis from the randomized evaluation of long-term anticoagulant therapy study. Circulation. 2013 Nov 12;128(20):2192-201. doi: 10.1161/CIRCULATIONAHA.112.000491. Epub 2013 Sep 9. PMID 24016454
- [Derived] Eikelboom JW, Connolly SJ, Hart RG, Wallentin L, Reilly P, Oldgren J, Yang S, Yusuf S. Balancing the benefits and risks of 2 doses of dabigatran compared with warfarin in atrial fibrillation. J Am Coll Cardiol. 2013 Sep 3;62(10):900-8. doi: 10.1016/j.jacc.2013.05.042. Epub 2013 Jun 13. PMID 23770182
- [Derived] Hori M, Connolly SJ, Zhu J, Liu LS, Lau CP, Pais P, Xavier D, Kim SS, Omar R, Dans AL, Tan RS, Chen JH, Tanomsup S, Watanabe M, Koyanagi M, Ezekowitz MD, Reilly PA, Wallentin L, Yusuf S; RE-LY Investigators. Dabigatran versus warfarin: effects on ischemic and hemorrhagic strokes and bleeding in Asians and non-Asians with atrial fibrillation. Stroke. 2013 Jul;44(7):1891-6. doi: 10.1161/STROKEAHA.113.000990. Epub 2013 Jun 6. PMID 23743976
- [Derived] Pare G, Eriksson N, Lehr T, Connolly S, Eikelboom J, Ezekowitz MD, Axelsson T, Haertter S, Oldgren J, Reilly P, Siegbahn A, Syvanen AC, Wadelius C, Wadelius M, Zimdahl-Gelling H, Yusuf S, Wallentin L. Genetic determinants of dabigatran plasma levels and their relation to bleeding. Circulation. 2013 Apr 2;127(13):1404-12. doi: 10.1161/CIRCULATIONAHA.112.001233. Epub 2013 Mar 6. PMID 23467860
- [Derived] Dans AL, Connolly SJ, Wallentin L, Yang S, Nakamya J, Brueckmann M, Ezekowitz M, Oldgren J, Eikelboom JW, Reilly PA, Yusuf S. Concomitant use of antiplatelet therapy with dabigatran or warfarin in the Randomized Evaluation of Long-Term Anticoagulation Therapy (RE-LY) trial. Circulation. 2013 Feb 5;127(5):634-40. doi: 10.1161/CIRCULATIONAHA.112.115386. Epub 2012 Dec 27. PMID 23271794
- [Derived] Bytzer P, Connolly SJ, Yang S, Ezekowitz M, Formella S, Reilly PA, Aisenberg J. Analysis of upper gastrointestinal adverse events among patients given dabigatran in the RE-LY trial. Clin Gastroenterol Hepatol. 2013 Mar;11(3):246-52.e1-5. doi: 10.1016/j.cgh.2012.10.021. Epub 2012 Oct 24. PMID 23103906
- [Derived] Van Spall HG, Wallentin L, Yusuf S, Eikelboom JW, Nieuwlaat R, Yang S, Kabali C, Reilly PA, Ezekowitz MD, Connolly SJ. Variation in warfarin dose adjustment practice is responsible for differences in the quality of anticoagulation control between centers and countries: an analysis of patients receiving warfarin in the randomized evaluation of long-term anticoagulation therapy (RE-LY) trial. Circulation. 2012 Nov 6;126(19):2309-16. doi: 10.1161/CIRCULATIONAHA.112.101808. Epub 2012 Oct 1. PMID 23027801
- [Derived] Healey JS, Eikelboom J, Douketis J, Wallentin L, Oldgren J, Yang S, Themeles E, Heidbuchel H, Avezum A, Reilly P, Connolly SJ, Yusuf S, Ezekowitz M; RE-LY Investigators. Periprocedural bleeding and thromboembolic events with dabigatran compared with warfarin: results from the Randomized Evaluation of Long-Term Anticoagulation Therapy (RE-LY) randomized trial. Circulation. 2012 Jul 17;126(3):343-8. doi: 10.1161/CIRCULATIONAHA.111.090464. Epub 2012 Jun 14. PMID 22700854
- [Derived] Hijazi Z, Oldgren J, Andersson U, Connolly SJ, Ezekowitz MD, Hohnloser SH, Reilly PA, Vinereanu D, Siegbahn A, Yusuf S, Wallentin L. Cardiac biomarkers are associated with an increased risk of stroke and death in patients with atrial fibrillation: a Randomized Evaluation of Long-term Anticoagulation Therapy (RE-LY) substudy. Circulation. 2012 Apr 3;125(13):1605-16. doi: 10.1161/CIRCULATIONAHA.111.038729. Epub 2012 Feb 28. PMID 22374183
- [Derived] Hohnloser SH, Oldgren J, Yang S, Wallentin L, Ezekowitz M, Reilly P, Eikelboom J, Brueckmann M, Yusuf S, Connolly SJ. Myocardial ischemic events in patients with atrial fibrillation treated with dabigatran or warfarin in the RE-LY (Randomized Evaluation of Long-Term Anticoagulation Therapy) trial. Circulation. 2012 Feb 7;125(5):669-76. doi: 10.1161/CIRCULATIONAHA.111.055970. Epub 2012 Jan 3. PMID 22215856
- [Derived] Oldgren J, Alings M, Darius H, Diener HC, Eikelboom J, Ezekowitz MD, Kamensky G, Reilly PA, Yang S, Yusuf S, Wallentin L, Connolly SJ; RE-LY Investigators. Risks for stroke, bleeding, and death in patients with atrial fibrillation receiving dabigatran or warfarin in relation to the CHADS2 score: a subgroup analysis of the RE-LY trial. Ann Intern Med. 2011 Nov 15;155(10):660-7, W204. doi: 10.7326/0003-4819-155-10-201111150-00004. PMID 22084332
- [Derived] Eikelboom JW, Wallentin L, Connolly SJ, Ezekowitz M, Healey JS, Oldgren J, Yang S, Alings M, Kaatz S, Hohnloser SH, Diener HC, Franzosi MG, Huber K, Reilly P, Varrone J, Yusuf S. Risk of bleeding with 2 doses of dabigatran compared with warfarin in older and younger patients with atrial fibrillation: an analysis of the randomized evaluation of long-term anticoagulant therapy (RE-LY) trial. Circulation. 2011 May 31;123(21):2363-72. doi: 10.1161/CIRCULATIONAHA.110.004747. Epub 2011 May 16. PMID 21576658
- [Derived] Nagarakanti R, Ezekowitz MD, Oldgren J, Yang S, Chernick M, Aikens TH, Flaker G, Brugada J, Kamensky G, Parekh A, Reilly PA, Yusuf S, Connolly SJ. Dabigatran versus warfarin in patients with atrial fibrillation: an analysis of patients undergoing cardioversion. Circulation. 2011 Jan 18;123(2):131-6. doi: 10.1161/CIRCULATIONAHA.110.977546. Epub 2011 Jan 3. PMID 21200007
- [Derived] Ezekowitz MD, Wallentin L, Connolly SJ, Parekh A, Chernick MR, Pogue J, Aikens TH, Yang S, Reilly PA, Lip GY, Yusuf S; RE-LY Steering Committee and Investigators. Dabigatran and warfarin in vitamin K antagonist-naive and -experienced cohorts with atrial fibrillation. Circulation. 2010 Nov 30;122(22):2246-53. doi: 10.1161/CIRCULATIONAHA.110.973735. PMID 21147728
- [Derived] Diener HC, Connolly SJ, Ezekowitz MD, Wallentin L, Reilly PA, Yang S, Xavier D, Di Pasquale G, Yusuf S; RE-LY study group. Dabigatran compared with warfarin in patients with atrial fibrillation and previous transient ischaemic attack or stroke: a subgroup analysis of the RE-LY trial. Lancet Neurol. 2010 Dec;9(12):1157-1163. doi: 10.1016/S1474-4422(10)70274-X. Epub 2010 Nov 6. PMID 21059484
- [Derived] Wallentin L, Yusuf S, Ezekowitz MD, Alings M, Flather M, Franzosi MG, Pais P, Dans A, Eikelboom J, Oldgren J, Pogue J, Reilly PA, Yang S, Connolly SJ; RE-LY investigators. Efficacy and safety of dabigatran compared with warfarin at different levels of international normalised ratio control for stroke prevention in atrial fibrillation: an analysis of the RE-LY trial. Lancet. 2010 Sep 18;376(9745):975-83. doi: 10.1016/S0140-6736(10)61194-4. PMID 20801496
- [Derived] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Derived] Ezekowitz MD, Connolly S, Parekh A, Reilly PA, Varrone J, Wang S, Oldgren J, Themeles E, Wallentin L, Yusuf S. Rationale and design of RE-LY: randomized evaluation of long-term anticoagulant therapy, warfarin, compared with dabigatran. Am Heart J. 2009 May;157(5):805-10, 810.e1-2. doi: 10.1016/j.ahj.2009.02.005. PMID 19376304

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran 110 mg: 110 mg twice daily, total daily dose 220 mg
- Dabigatran 150 mg: 150 mg twice daily, total daily dose 300 mg
- Warfarin: Target International Normalized Ratio (INR) of 2.0 to 3.0
Period: Overall Study
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Started | 6015 | 6076 | 6022
Completed | 5780 | 5824 | 5756
Not Completed | 235 | 252 | 266
Not completed — Lost to Follow-up | 17 | 31 | 41
Not completed — Withdrawal by Subject | 128 | 145 | 139
Not completed — Not Treated | 32 | 17 | 24
Not completed — Other | 58 | 59 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin | Total
Number analyzed (Participants) | 6015 | 6076 | 6022 | 18113
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (8.6) | 71.5 (8.8) | 71.6 (8.6) | 71.5 (8.7)
Age, Customized [Number; unit: Participants]
  <65 | 998 | 1030 | 953 | 2981
  65<= and <75 | 2668 | 2580 | 2646 | 7894
  >=75 | 2349 | 2466 | 2423 | 7238
Sex/Gender, Customized [Number; unit: participants]
  Male | 3865 | 3840 | 3809 | 11514
  Female | 2149 | 2236 | 2213 | 6598
  Missing | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 5593 | 5660 | 5615 | 16868
  Hispanic or Latino | 421 | 416 | 407 | 1244
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4208 | 4268 | 4203 | 12679
  Black | 52 | 57 | 67 | 176
  Asian | 955 | 965 | 955 | 2875
  Other | 799 | 786 | 797 | 2382
  Missing | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  USA, Canada | 2166 | 2200 | 2167 | 6533
  Central Europe | 707 | 706 | 706 | 2119
  Western Europe | 1544 | 1555 | 1552 | 4651
  Latin America | 320 | 320 | 316 | 956
  Asia | 923 | 933 | 926 | 2782
  Other | 355 | 362 | 355 | 1072
Smoking history [Number; unit: participants]
  Non-smoker | 2941 | 2993 | 3006 | 8940
  Smoker | 440 | 447 | 448 | 1335
  Ex-smoker | 2633 | 2636 | 2567 | 7836
  Missing | 1 | 0 | 1 | 2
Regular Alcohol Consumption [Number; unit: participants]
  No | 4017 | 4077 | 4040 | 12134
  Yes | 1996 | 1999 | 1981 | 5976
  Missing | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Yearly Event Rate for Composite Endpoint of Stroke/SEE
Description: Time to first occurrence of stroke or systemic embolic event. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum(date of study termination - date of randomization + 1) of all randomized subjects / 365.25
Time Frame: 36 months
Population: Randomized set - The randomized set includes all randomized subjects in the treatment groups to which they were randomized, regardless of whether the subjects took randomized study medication or not.
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 6015 | 6076 | 6022
yearly event rate (percentage) | 1.54 | 1.11 | 1.71
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Warfarin; Non-inferiority comparison of dabigatran 110 mg to warfarin; Test type: Non-Inferiority or Equivalence — Comparisons between treatment groups were performed using a Cox regression analysis with treatment in the model; p < .0001, Regression, Cox — p-value for protocol specified margin of 1.46; Cox Proportional Hazard = 0.90, 95% CI [0.74 to 1.10]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Non-inferiority comparison of dabigatran 150 mg to warfarin; Test type: Non-Inferiority or Equivalence — Comparisons between treatment groups were performed using a Cox regression analysis with treatment in the model; p < .0001, Regression, Cox — p-value for protocol specified margin of 1.46; Cox Proportional Hazard = 0.65, 95% CI [0.52 to 0.81]

2. Secondary Outcome: Yearly Event Rate for Composite Endpoint of Stroke/SEE/All Cause Death
Description: Time to first occurrence of stroke, SEE or all cause death. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum(date of study termination - date of randomization + 1) of all randomized subjects / 365.25
Time Frame: 36 months
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 6015 | 6076 | 6022
yearly event rate (percentage) | 4.85 | 4.32 | 5.20
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Warfarin; Test type: Superiority or Other; p = 0.2206, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using a Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.93, 95% CI [0.83 to 1.04]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Test type: Superiority or Other; p = 0.0015, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using a Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.83, 95% CI [0.74 to 0.93]

3. Secondary Outcome: Yearly Event Rate: Composite of Stroke/SEE/PE/MI/Vascular Death
Description: Time to first occurrence of stroke, systemic embolic event, pulmonary embolism, myocardial infarction including silent myocardial infarction or vascular death. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum(date of study termination - date of randomization + 1) of all randomized subjects / 365.25
Time Frame: 36 months
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 6015 | 6076 | 6022
yearly event rate (percentage) | 4.26 | 3.68 | 4.35
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Warfarin; Test type: Superiority or Other; p = 0.7508, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using a Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.98, 95% CI [0.87 to 1.11]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Test type: Superiority or Other; p = 0.0093, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using a Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.84, 95% CI [0.74 to 0.96]

4. Secondary Outcome: Bleeding Events (Major and Minor)
Description: Yearly event rate of bleeds. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum(date of study termination - date of randomization + 1) of all randomized subjects / 365.25
  Major bleeds are adjudicated, whereas minor bleeds are investigator reported.
Time Frame: 36 months
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 6015 | 6076 | 6022
yearly event rate (percentage)
  Major bleeds | 2.99 | 3.55 | 3.81
  Minor bleeds | 13.16 | 14.85 | 16.37
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Warfarin; Analysis is for adjudicated major bleeds; Test type: Superiority or Other; p = 0.0026, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.80, 95% CI [0.70 to 0.93]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Analysis is for adjudicated major bleeds; Test type: Superiority or Other; p = 0.3146, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.93, 95% CI [0.81 to 1.07]

5. Secondary Outcome: Clinical Relevant Abnormalities for Intracerebral Hemorrhage and Other Intracranial Hemorrhage (ICH)
Description: Patients with clinical relevant abnormalities for intracerebral hemorrhage, other intracranial hemorrhage (ICH)
Time Frame: 36 months
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)]
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 5983 | 6059 | 5998
yearly event rate (percentage)]
  intracerebral hemorrhage | 0.12 | 0.10 | 0.38
  intracranial hemorrhage (ICH) | 0.23 | 0.32 | 0.76
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Warfarin; Analysis of ICH; Test type: Superiority or Other; p < 0.0001, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.30, 95% CI [0.19 to 0.45]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Analysis of ICH; Test type: Superiority or Other; p < 0.0001, Regression, Cox — p-value is for superiority testing; Comparisons between treatment groups were performed using Cox regression analysis with treatment in the model; Cox Proportional Hazard = 0.41, 95% CI [0.28 to 0.60]

6. Secondary Outcome: Abnormal Liver Function Test
Description: Number of subjects with abnormal liver function test (LFT), i.e., ALT/AST>3xULN and total bilirubin > 2 x ULN
Time Frame: 36 months
Population: Safety set - all subjects who were randomized and received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 5983 | 6059 | 5998
participants | 11 | 14 | 21

ADVERSE EVENTS:
Time Frame: 36 months
Description: Number of participants at risk represents the number of participants who received study medication. The following number of subjects did not take any study drug after randomization: 32 assigned to Dabigatran 110 mg; 17 assigned to Dabigatran 150 mg; and 24 assigned to Warfarin.
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Warfarin
Serious Adverse Events (participants affected / at risk) | 1263/5983 | 1289/6059 | 1357/5998
Other Adverse Events (participants affected / at risk) | 2286/5983 | 2273/6059 | 2118/5998
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 110 mg (N=5983) | Dabigatran 150 mg (N=6059) | Warfarin (N=5998)
Anaemia (Blood and lymphatic system disorders) | 34 | 47 | 33
Coagulopathy (Blood and lymphatic system disorders) | 4 | 3 | 12
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 6 | 5 | 10
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2 | 3
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 | 1 | 0
Lymphatic disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 3 | 1
Sideroblastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 6 | 3
Acute coronary syndrome (Cardiac disorders) | 5 | 8 | 4
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 4
Angina pectoris (Cardiac disorders) | 29 | 30 | 22
Angina unstable (Cardiac disorders) | 7 | 13 | 5
Aortic valve calcification (Cardiac disorders) | 0 | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 2 | 0 | 3
Aortic valve sclerosis (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 4 | 2 | 1
Arrhythmia (Cardiac disorders) | 6 | 1 | 4
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 64 | 55 | 74
Atrial flutter (Cardiac disorders) | 5 | 10 | 5
Atrial thrombosis (Cardiac disorders) | 7 | 5 | 1
Atrioventricular block (Cardiac disorders) | 2 | 2 | 2
Atrioventricular block complete (Cardiac disorders) | 2 | 4 | 5
Atrioventricular block first degree (Cardiac disorders) | 3 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 20 | 21 | 20
Cardiac arrest (Cardiac disorders) | 8 | 5 | 5
Cardiac asthma (Cardiac disorders) | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 51 | 62 | 65
Cardiac failure acute (Cardiac disorders) | 5 | 1 | 7
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 83 | 58 | 73
Cardiac perforation (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2 | 2
Cardiogenic shock (Cardiac disorders) | 4 | 1 | 6
Cardiomegaly (Cardiac disorders) | 1 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Cor pulmonale (Cardiac disorders) | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 9 | 10 | 11
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Coronary artery perforation (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 2
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 2 | 0 | 2
Left ventricular failure (Cardiac disorders) | 1 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 6 | 4 | 10
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 2 | 1
Nodal rhythm (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 7 | 2 | 5
Pericardial effusion (Cardiac disorders) | 4 | 4 | 5
Pericardial haemorrhage (Cardiac disorders) | 1 | 3 | 3
Pericarditis (Cardiac disorders) | 1 | 1 | 2
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 3
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 2
Sick sinus syndrome (Cardiac disorders) | 8 | 3 | 8
Sinoatrial block (Cardiac disorders) | 0 | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 5
Torsade de pointes (Cardiac disorders) | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 2 | 1 | 5
Ventricular arrhythmia (Cardiac disorders) | 5 | 5 | 3
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 3 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 6 | 3 | 10
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 1 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 1
Congenital arterial malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 0 | 0 | 1
Exomphalos (Congenital, familial and genetic disorders) | 0 | 2 | 0
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 2 | 0 | 0
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1 | 2 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 2 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0
External ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 5 | 6 | 14
Vertigo positional (Ear and labyrinth disorders) | 3 | 2 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 2 | 0
Addison's disease (Endocrine disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0 | 1
Goitre (Endocrine disorders) | 0 | 5 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 3 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 3 | 2
Hypothyroidism (Endocrine disorders) | 2 | 1 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Thyrotoxic crisis (Endocrine disorders) | 0 | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 1 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 7 | 6 | 11
Conjunctival discolouration (Eye disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 1
Diabetic retinopathy (Eye disorders) | 2 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 4 | 3 | 6
Glaucoma (Eye disorders) | 2 | 1 | 0
Hyphaema (Eye disorders) | 2 | 2 | 0
Hypotony of eye (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1
Macular degeneration (Eye disorders) | 3 | 1 | 0
Necrotising retinitis (Eye disorders) | 0 | 1 | 0
Optic neuropathy (Eye disorders) | 0 | 0 | 1
Pseudophakia (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 3 | 1 | 3
Retinal haemorrhage (Eye disorders) | 3 | 1 | 1
Retinal tear (Eye disorders) | 1 | 0 | 0
Retinitis (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 2 | 0 | 1
Visual impairment (Eye disorders) | 1 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 3 | 3 | 3
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 8 | 17
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5 | 4
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Anal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 3 | 3 | 3
Coeliac disease (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 3 | 2 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 2 | 5
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 4
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 7 | 20
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 1 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 2 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 3 | 4 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Dyskinesia oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 6 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 3 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Enterocele (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 2 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 5 | 5 | 4
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 5 | 5
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 6 | 6 | 6
Gastritis erosive (Gastrointestinal disorders) | 5 | 4 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 | 3 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 38 | 55 | 41
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 4 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 3 | 3
Haematemesis (Gastrointestinal disorders) | 2 | 5 | 2
Haematochezia (Gastrointestinal disorders) | 5 | 2 | 3
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 3 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 3 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 1 | 1
Hiatus hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 8 | 1 | 2
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 15 | 16 | 12
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 2
Intestinal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 2 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 2 | 4
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 2
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 1 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 12 | 3
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 | 1 | 0
Melaena (Gastrointestinal disorders) | 7 | 10 | 6
Melanosis coli (Gastrointestinal disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 7 | 9
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal mass (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 2 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 4 | 8
Pancreatitis acute (Gastrointestinal disorders) | 3 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 2 | 0 | 2
Peritoneal cyst (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 3
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0
Presbyoesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 15 | 13 | 9
Rectal lesion (Gastrointestinal disorders) | 1 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Salivary gland cyst (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 4 | 2
Stress ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 13 | 12
Volvulus (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 17 | 6 | 9
Adhesion (General disorders) | 0 | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0 | 3
Asthenia (General disorders) | 12 | 10 | 15
Chest discomfort (General disorders) | 3 | 4 | 2
Chest pain (General disorders) | 29 | 45 | 46
Chills (General disorders) | 0 | 0 | 1
Condition aggravated (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 1 | 0 | 0
Death (General disorders) | 4 | 4 | 0
Discomfort (General disorders) | 1 | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 6 | 12
Feeling abnormal (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 3 | 2
General physical health deterioration (General disorders) | 1 | 3 | 5
Generalised oedema (General disorders) | 0 | 0 | 1
Hernia (General disorders) | 2 | 2 | 2
Hernia obstructive (General disorders) | 1 | 1 | 0
Hyperthermia (General disorders) | 2 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 1
Implant site inflammation (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1
Ischaemic ulcer (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 2 | 0
Mass (General disorders) | 1 | 0 | 0
Mechanical complication of implant (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 5 | 3 | 6
Necrosis (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 3 | 5
Oedema (General disorders) | 2 | 1 | 3
Oedema peripheral (General disorders) | 10 | 3 | 13
Pain (General disorders) | 1 | 2 | 6
Pelvic mass (General disorders) | 1 | 0 | 1
Polyp (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 11 | 13 | 14
Sudden cardiac death (General disorders) | 2 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 1
Ulcer (General disorders) | 0 | 1 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 2 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 8 | 8 | 9
Cholecystitis acute (Hepatobiliary disorders) | 4 | 3 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 7 | 3 | 7
Cholestasis (Hepatobiliary disorders) | 0 | 2 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 3 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 2 | 0
Amyloidosis (Immune system disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Primary amyloidosis (Immune system disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 1
Abscess intestinal (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 3 | 2 | 4
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 4 | 2 | 2
Appendiceal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 5 | 11 | 7
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 2 | 2 | 2
Arthritis infective (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 4 | 2 | 2
Bacterial sepsis (Infections and infestations) | 3 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 11 | 13 | 11
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 2 | 3
Bursitis infective (Infections and infestations) | 0 | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0 | 0
Catheter sepsis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 21 | 23 | 20
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Cervicitis (Infections and infestations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 2 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 3 | 1 | 1
Creutzfeldt-Jakob disease (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 2 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 2 | 3 | 4
Diabetic gangrene (Infections and infestations) | 0 | 2 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 5 | 5 | 12
Empyema (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 3 | 3 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 4 | 7 | 3
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 3 | 0 | 2
Eye infection viral (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 3 | 4 | 3
Gastroenteritis (Infections and infestations) | 11 | 13 | 8
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 3 | 3 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Helminthic infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 5 | 1
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0 | 0
Histoplasmosis (Infections and infestations) | 1 | 0 | 0
Implant site cellulitis (Infections and infestations) | 1 | 0 | 0
Implant site infection (Infections and infestations) | 1 | 3 | 2
Incision site cellulitis (Infections and infestations) | 0 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 2 | 1 | 1
Infection (Infections and infestations) | 0 | 3 | 3
Influenza (Infections and infestations) | 2 | 1 | 2
Infusion site infection (Infections and infestations) | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 3 | 0 | 1
Intestinal gangrene (Infections and infestations) | 0 | 1 | 0
Jejunal gangrene (Infections and infestations) | 0 | 0 | 1
Keratitis herpetic (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 6 | 3 | 5
Localised infection (Infections and infestations) | 3 | 4 | 3
Lower respiratory tract infection (Infections and infestations) | 3 | 1 | 3
Lung infection (Infections and infestations) | 2 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 4 | 8 | 2
Osteomyelitis acute (Infections and infestations) | 0 | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 2
Osteomyelitis salmonella (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 1
Peridiverticular abscess (Infections and infestations) | 0 | 0 | 1
Periorbital abscess (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 2 | 1
Peritoneal infection (Infections and infestations) | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 74 | 70 | 62
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 2
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 2 | 1
Postoperative abscess (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 5 | 0 | 1
Proteus infection (Infections and infestations) | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 2 | 0
Pyelonephritis (Infections and infestations) | 5 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 3 | 1 | 0
Pyonephrosis (Infections and infestations) | 1 | 0 | 0
Pyothorax (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Salmonella bacteraemia (Infections and infestations) | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 19 | 17 | 19
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 10 | 6 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 2 | 5 | 3
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Subacute endocarditis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 0
Superinfection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 2
Toxoplasmosis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 6
Urinary tract infection (Infections and infestations) | 18 | 13 | 21
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 10 | 4 | 4
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 3 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
West Nile viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 4 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1 | 5
Adrenal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Agitation postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 1 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Bladder injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 2 | 2 | 2
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1 | 0
Complication of device insertion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 3 | 5 | 2
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 1 | 4
Device breakage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Device dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device electrical finding (Injury, poisoning and procedural complications) | 1 | 2 | 0
Device failure (Injury, poisoning and procedural complications) | 0 | 2 | 4
Device lead damage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Drug administration error (Injury, poisoning and procedural complications) | 0 | 2 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Failure to capture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 22 | 29 | 43
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 4 | 8 | 6
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Flail chest (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 4 | 3 | 6
Heart injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 8 | 8 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1 | 2
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 2 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 1 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Lung injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 3 | 3 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nerve root injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 3 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 8
Pacemaker complication (Injury, poisoning and procedural complications) | 2 | 0 | 0
Pancreatic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Pocket erosion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 2 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 5 | 3
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 1 | 0 | 2
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 1 | 0
Retinal scar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 5 | 6 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 5 | 4
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 3 | 8 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 1 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Splenic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 4 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 3 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 5 | 11 | 20
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 6 | 5 | 9
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transurethral resection syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 2
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Underdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ventriculoperitoneal shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vertebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 2
Arteriogram coronary (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Biopsy (Investigations) | 1 | 0 | 0
Biopsy breast (Investigations) | 0 | 1 | 0
Biopsy endometrium (Investigations) | 0 | 0 | 1
Biopsy lung (Investigations) | 1 | 0 | 0
Biopsy prostate (Investigations) | 0 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 5 | 0
Blood glucose increased (Investigations) | 1 | 0 | 2
Blood osmolarity decreased (Investigations) | 0 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 1 | 0 | 3
Brain natriuretic peptide increased (Investigations) | 2 | 0 | 0
Carbohydrate antigen 125 increased (Investigations) | 1 | 0 | 0
Cardiac electrophysiologic study (Investigations) | 1 | 2 | 1
Cardiac stress test (Investigations) | 0 | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 0 | 1
Catheterisation cardiac (Investigations) | 1 | 0 | 5
Chest X-ray abnormal (Investigations) | 0 | 1 | 0
Coagulation factor increased (Investigations) | 1 | 0 | 0
Coagulation test abnormal (Investigations) | 0 | 1 | 1
Coagulation time prolonged (Investigations) | 0 | 0 | 3
Colonoscopy (Investigations) | 0 | 0 | 1
Colonoscopy abnormal (Investigations) | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 3 | 0
Echocardiogram abnormal (Investigations) | 1 | 0 | 0
Electroencephalogram abnormal (Investigations) | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 3 | 4
Haemoglobin decreased (Investigations) | 7 | 12 | 10
Heart rate increased (Investigations) | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 4 | 2
International normalised ratio increased (Investigations) | 0 | 1 | 19
Intraocular pressure increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 5 | 8 | 5
Lymphocyte count increased (Investigations) | 0 | 0 | 1
Megakaryocytes decreased (Investigations) | 1 | 0 | 0
Occult blood positive (Investigations) | 1 | 1 | 0
Oesophagogastroduodenoscopy (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0
Precancerous cells present (Investigations) | 0 | 1 | 0
Prostatic specific antigen (Investigations) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 1
Sinus rhythm (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Tumour marker increased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 1
Venous pressure jugular increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 6 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 15 | 22 | 31
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 6 | 7
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 5 | 3
Diabetic foot (Metabolism and nutrition disorders) | 4 | 3 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 3 | 3 | 7
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 18 | 4 | 12
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 11 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 5 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 9 | 10
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Ketosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Starvation (Metabolism and nutrition disorders) | 0 | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Articular disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 17 | 9
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 1 | 3
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 9 | 4 | 4
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 22 | 13 | 21
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Shoulder deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 13 | 14
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 3
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 17 | 10
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 3
Cardiac fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cardiac neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 17 | 8
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gallbladder cancer non-resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Gastric cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Inflammatory myofibroblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Langerhans' cell granulomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 2
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leiomyosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Leukaemia monocytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 3
Lung carcinoma cell type unspecified stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 8 | 14
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4 | 2
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 3
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 4
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 3
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 3
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 7
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 | 32 | 29
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 5
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 4
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 15 | 10
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8 | 2
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Urethral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 3
Amnesia (Nervous system disorders) | 0 | 1 | 2
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 1
Anoxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 1 | 1
Basilar artery occlusion (Nervous system disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Carotid artery disease (Nervous system disorders) | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 7 | 5
Carotid artery thrombosis (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1 | 0
Cerebral circulatory failure (Nervous system disorders) | 1 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 2 | 13
Cerebral hypoperfusion (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 3 | 3 | 2
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 7 | 1 | 5
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 2 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 2 | 2 | 0
Coma (Nervous system disorders) | 1 | 1 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 3 | 3
Dementia (Nervous system disorders) | 1 | 2 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 15 | 18 | 18
Dysarthria (Nervous system disorders) | 0 | 3 | 2
Embolic stroke (Nervous system disorders) | 1 | 0 | 1
Encephalitis (Nervous system disorders) | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 4 | 3 | 6
Epilepsy (Nervous system disorders) | 2 | 3 | 0
Facial palsy (Nervous system disorders) | 1 | 0 | 1
Frontotemporal dementia (Nervous system disorders) | 1 | 0 | 0
Global amnesia (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 1 | 5
Haemorrhagic stroke (Nervous system disorders) | 1 | 2 | 9
Headache (Nervous system disorders) | 1 | 4 | 3
Hemiparesis (Nervous system disorders) | 2 | 1 | 3
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0 | 0
Hypoxic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 2 | 1
Lacunar infarction (Nervous system disorders) | 2 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 2 | 0
Loss of consciousness (Nervous system disorders) | 3 | 4 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0
Narcolepsy (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neuritis (Nervous system disorders) | 0 | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 2 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 1
Paralysis (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 1 | 0
Peripheral paralysis (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Post-traumatic headache (Nervous system disorders) | 1 | 0 | 0
Posterior interosseous syndrome (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 3 | 7 | 5
Pseudoparalysis (Nervous system disorders) | 0 | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1 | 2
Subdural hygroma (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 33 | 31 | 34
Tension headache (Nervous system disorders) | 0 | 2 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 2 | 3
Tremor (Nervous system disorders) | 2 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 1
Wernicke's encephalopathy (Nervous system disorders) | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Apathy (Psychiatric disorders) | 1 | 0 | 0
Bereavement reaction (Psychiatric disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 7 | 8 | 10
Delirium (Psychiatric disorders) | 1 | 2 | 4
Delusion (Psychiatric disorders) | 0 | 1 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 6 | 8 | 6
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 2 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 1
Mania (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 4 | 9 | 6
Panic attack (Psychiatric disorders) | 1 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1 | 0
Somatisation disorder (Psychiatric disorders) | 1 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 1
Withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 2 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 1
Bladder mass (Renal and urinary disorders) | 0 | 2 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 0 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 2 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 4 | 1 | 3
Calculus urinary (Renal and urinary disorders) | 1 | 1 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 16 | 14 | 15
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 3 | 0 | 2
Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 5 | 3 | 8
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Nephrosclerosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 2 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 2 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 1 | 2
Renal colic (Renal and urinary disorders) | 0 | 0 | 2
Renal cyst (Renal and urinary disorders) | 0 | 1 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 15 | 19 | 27
Renal failure acute (Renal and urinary disorders) | 42 | 38 | 35
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 2
Renal impairment (Renal and urinary disorders) | 3 | 5 | 2
Renal mass (Renal and urinary disorders) | 3 | 3 | 4
Renal pain (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 3 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 4 | 1 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 1 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 6 | 4 | 6
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 7 | 5 | 5
Breast mass (Reproductive system and breast disorders) | 0 | 2 | 2
Colpocele (Reproductive system and breast disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 2
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 2
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 3
Prostatic disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 3 | 3 | 2
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal haematocoele (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1 | 2
Vaginal disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 2 | 1
Vaginal polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 2 | 1 | 0
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 8
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 24 | 14 | 20
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Diaphragmatic rupture (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 | 43 | 45
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Eosinophilic pneumonia acute (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 17
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 9
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 22 | 17 | 21
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 9
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 15
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Campbell de Morgan spots (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Photosensitivity allergic reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 4 | 6
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Joint prosthesis user (Social circumstances) | 1 | 0 | 0
Refusal of treatment by patient (Social circumstances) | 0 | 0 | 1
Walking disability (Social circumstances) | 1 | 0 | 0
Alcohol rehabilitation (Surgical and medical procedures) | 1 | 1 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 2 | 0 | 0
Aortic valve repair (Surgical and medical procedures) | 0 | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 0 | 2
Arthrodesis (Surgical and medical procedures) | 0 | 0 | 1
Artificial urinary sphincter implant (Surgical and medical procedures) | 0 | 0 | 1
Bladder neoplasm surgery (Surgical and medical procedures) | 1 | 0 | 0
Bladder operation (Surgical and medical procedures) | 1 | 0 | 0
Cardiac ablation (Surgical and medical procedures) | 1 | 0 | 1
Cardiac operation (Surgical and medical procedures) | 0 | 0 | 1
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 9 | 7 | 10
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 3 | 1
Cardiac pacemaker revision (Surgical and medical procedures) | 0 | 1 | 1
Cardioversion (Surgical and medical procedures) | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 2 | 0 | 1
Chemotherapy (Surgical and medical procedures) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 2
Colon operation (Surgical and medical procedures) | 1 | 0 | 0
Contraceptive diaphragm (Surgical and medical procedures) | 0 | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 1 | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 0 | 2 | 2
Craniotomy (Surgical and medical procedures) | 0 | 0 | 1
Debridement (Surgical and medical procedures) | 1 | 0 | 0
Dupuytren's contracture operation (Surgical and medical procedures) | 1 | 0 | 0
Endarterectomy (Surgical and medical procedures) | 1 | 0 | 0
Eventration procedure (Surgical and medical procedures) | 0 | 1 | 0
Explorative laparotomy (Surgical and medical procedures) | 1 | 0 | 0
Eye operation (Surgical and medical procedures) | 0 | 0 | 1
Gamma radiation therapy to prostate (Surgical and medical procedures) | 0 | 1 | 0
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 | 0 | 0
Heart valve operation (Surgical and medical procedures) | 1 | 0 | 0
Hepatectomy (Surgical and medical procedures) | 0 | 0 | 1
Hernia repair (Surgical and medical procedures) | 0 | 0 | 1
High frequency ablation (Surgical and medical procedures) | 2 | 2 | 1
Hip arthroplasty (Surgical and medical procedures) | 2 | 3 | 5
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 1
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 | 0 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 2 | 1 | 3
Incisional hernia repair (Surgical and medical procedures) | 0 | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 1 | 0
Internal fixation of fracture (Surgical and medical procedures) | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 1
Laparoscopic surgery (Surgical and medical procedures) | 0 | 0 | 1
Malignant tumour excision (Surgical and medical procedures) | 1 | 0 | 0
Mass excision (Surgical and medical procedures) | 0 | 1 | 0
Mastectomy (Surgical and medical procedures) | 1 | 1 | 0
Medical device implantation (Surgical and medical procedures) | 1 | 0 | 0
Medical device removal (Surgical and medical procedures) | 1 | 0 | 0
Mitral valve repair (Surgical and medical procedures) | 0 | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 0 | 0 | 1
Nerve block (Surgical and medical procedures) | 0 | 0 | 1
Open reduction of fracture (Surgical and medical procedures) | 1 | 0 | 1
Osteosynthesis (Surgical and medical procedures) | 1 | 0 | 0
Patellectomy (Surgical and medical procedures) | 1 | 0 | 0
Pleurodesis (Surgical and medical procedures) | 0 | 0 | 1
Polymedication (Surgical and medical procedures) | 1 | 0 | 0
Prostatic operation (Surgical and medical procedures) | 0 | 1 | 0
Radiotherapy (Surgical and medical procedures) | 1 | 1 | 0
Resuscitation (Surgical and medical procedures) | 0 | 0 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 0
Small intestinal resection (Surgical and medical procedures) | 0 | 0 | 1
Spinal laminectomy (Surgical and medical procedures) | 0 | 2 | 1
Stent placement (Surgical and medical procedures) | 1 | 0 | 1
Sternotomy (Surgical and medical procedures) | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 2 | 1 | 0
Tendon operation (Surgical and medical procedures) | 1 | 0 | 0
Thoracotomy (Surgical and medical procedures) | 3 | 0 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 0 | 1
Toe amputation (Surgical and medical procedures) | 1 | 0 | 0
Transfusion (Surgical and medical procedures) | 0 | 0 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 0 | 0 | 2
Umbilical hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 0 | 0 | 1
Wound drainage (Surgical and medical procedures) | 0 | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 0 | 1
Aneurysm (Vascular disorders) | 1 | 1 | 0
Angiodysplasia (Vascular disorders) | 0 | 2 | 0
Aortic aneurysm (Vascular disorders) | 8 | 8 | 9
Aortic aneurysm rupture (Vascular disorders) | 1 | 1 | 1
Aortic calcification (Vascular disorders) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 3 | 1 | 1
Aortic occlusion (Vascular disorders) | 0 | 1 | 0
Aortic rupture (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 11 | 5 | 8
Aortic thrombosis (Vascular disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 2 | 1 | 2
Arterial stenosis limb (Vascular disorders) | 0 | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 3 | 0 | 0
Arteriosclerosis (Vascular disorders) | 2 | 1 | 0
Arteriosclerosis obliterans (Vascular disorders) | 3 | 1 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 2 | 2
Deep vein thrombosis (Vascular disorders) | 7 | 4 | 4
Embolism (Vascular disorders) | 1 | 0 | 0
Exsanguination (Vascular disorders) | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 1 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 1 | 1
Haematoma (Vascular disorders) | 4 | 7 | 13
Haemorrhage (Vascular disorders) | 7 | 9 | 8
Hypertension (Vascular disorders) | 16 | 10 | 10
Hypertensive crisis (Vascular disorders) | 1 | 1 | 3
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 17 | 9 | 14
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 2 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 3 | 2 | 2
Ischaemia (Vascular disorders) | 0 | 0 | 1
Jugular vein distension (Vascular disorders) | 0 | 1 | 0
Leriche syndrome (Vascular disorders) | 0 | 0 | 1
Lymphangiectasia (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 4 | 4 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 3 | 4
Peripheral artery aneurysm (Vascular disorders) | 0 | 2 | 2
Peripheral embolism (Vascular disorders) | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 6 | 2
Peripheral vascular disorder (Vascular disorders) | 5 | 6 | 1
Phlebitis (Vascular disorders) | 1 | 1 | 0
Phlebitis deep (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 2 | 0
Subclavian artery thrombosis (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 2 | 1 | 0
Thrombosis (Vascular disorders) | 2 | 2 | 2
Varicose vein (Vascular disorders) | 2 | 0 | 1
Varicose vein ruptured (Vascular disorders) | 0 | 0 | 1
Vascular insufficiency (Vascular disorders) | 1 | 1 | 0
Vascular occlusion (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1
Venous haemorrhage (Vascular disorders) | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 2
Venous thrombosis limb (Vascular disorders) | 2 | 0 | 1
Wound haemorrhage (Vascular disorders) | 0 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 110 mg (N=5983) | Dabigatran 150 mg (N=6059) | Warfarin (N=5998)
Diarrhoea (Gastrointestinal disorders) | 347 | 360 | 308
Dyspepsia (Gastrointestinal disorders) | 362 | 344 | 83
Chest pain (General disorders) | 258 | 310 | 296
Fatigue (General disorders) | 367 | 361 | 341
Oedema peripheral (General disorders) | 436 | 439 | 440
Nasopharyngitis (Infections and infestations) | 315 | 309 | 327
Back pain (Musculoskeletal and connective tissue disorders) | 281 | 272 | 322
Dizziness (Nervous system disorders) | 442 | 440 | 536
Cough (Respiratory, thoracic and mediastinal disorders) | 318 | 308 | 343
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 460 | 483 | 506
Arthralgia (Musculoskeletal and connective tissue disorders) | 246 | 306 | 318

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.